CLINICAL TRIAL: NCT02045797
Title: A Phase II, Randomized, Two-Part, Multicenter, Dose-Ranging Study in Adult Subjects Evaluating the Safety, Tolerability, and Efficacy of GSK2140944 in the Treatment of Subjects With Suspected or Confirmed Gram-Positive Acute Bacterial Skin and Skin Structure Infections
Brief Title: Dose-Ranging Study of GSK2140944 in the Treatment of Subjects With Suspected or Confirmed Gram-Positive Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116704
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Infections, Bacterial
Keywords: Dose ranging; Intravenous; Adaptive design; suspected or confirmed gram-positive acute bacterial skin and skin structure infection; Subjects; infection; Oral; GSK2140944
MeSH Terms: conditions — Bacterial Infections; Infections | interventions — gepotidacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Group A (Experimental): Subject will receive GSK2140944 750mg IV every 12 hours (q12h; twice daily [BID]) on Day 1 and Day 2. Subject may switch to GSK2140944 1500mg orally (PO) q12h (BID) at investigator's decision or will continue to receive GSK2140944 750mg IV q12h (BID) from Day 3 to Day 10.
  Interventions: Drug: GSK2140944 Lyophile; Drug: GSK2140944 Capsules
- Treatment Group B (Experimental): Subject will receive GSK2140944 1000mg IV q12h (BID) on Day 1 and Day 2 . Subject may switch to GSK2140944 2000mg PO q12h (BID) at investigator's decision or will continue to receive GSK2140944 1000mg IV q12h (BID) from Day 3 to Day 10.
  Interventions: Drug: GSK2140944 Lyophile; Drug: GSK2140944 Capsules
- Treatment Group C (Experimental): Subject will receive GSK2140944 1000mg IV q8h (TID) on Day 1 and Day 2. Subject may switch to GSK2140944 2000mg PO q8h (TID) at investigator's decision or will continue to receive GSK2140944 1000mg IV q8h (TID) from Day 3 to Day 10.
  Interventions: Drug: GSK2140944 Lyophile; Drug: GSK2140944 Capsules

INTERVENTIONS:
Drug: GSK2140944 Lyophile — GSK2140944 Lyophile (pale yellow to grayish yellow cake) containing 750 mg of GSK2140944 (as free base) per vial for IV infusion.
Drug: GSK2140944 Capsules — GSK2140944 500 mg capsules will be supplied as pink hard gelatin capsule with no external markings filled with slightly agglomerated pale yellow to grayish yellow powder.

SUMMARY:
GSK2140944 belongs to a novel structural class of antibiotics - Bacterial Type II Topoisomerase Inhibitors (BTI). This is a Phase II, randomized, two-part, multicenter study designed to select the optimal dose by further characterizing the safety, tolerability and PK of GSK 2140944 and by evaluating efficacy in subjects requiring in-patient medical care to treat their suspected or confirmed Gram-positive acute bacterial skin and skin structure infections (ABSSSI). The selected dose will be used in future studies.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adult male at least 18 years of age or an adult female at least 18 years of age who meets one of the following criteria: A female of child-bearing potential who is either 1) sexually inactive by abstinence, 2) whose sole male partner has been sterilized, or 3) uses a contraceptive method with a failure rate of < 1%. Females of child-bearing potential must not become pregnant during the study. A female of non child- bearing potential, which includes: Females who are surgically sterile with a documented hysterectomy and/or bilateral oophorectomy; Females with a documented tubal ligation. If the procedure was done hysteroscopically, the effectiveness of tubal occlusion must have been documented by hysterosalpingogram post procedure (typically 3 months after procedure); Females who are post-menopausal, defined as amenorrhoeic for greater than 1 year. For women whose menopausal status is in doubt, a documented previous confirmatory blood sample with follicle-stimulating hormone (FSH) > 40 milli-international units per milliliter (MIU/mL) and estradiol <40 picograms per milliliter (<140 picomole per liter) would need to be confirmed or they will be required to use one of the contraception methods.
* The subject has a diagnosis of ABSSSI suspected or documented to be caused by Gram-positive pathogens that requires of intravenous (IV) antibiotic treatment for which subjects is willing to receive treatment in an in-patient setting for at least 2 days.. ABSSSI is defined as one of the following: Wound infection (traumatic or post-surgical): an infection involving skin and subcutaneous tissue, characterized by purulent drainage from a wound with surrounding redness, edema, and/or induration of a minimum surface area of 75 square centimeter (cm^2) (e.g., the shortest distance of redness, edema, and/or induration extending at least 5 centimeter (cm) from the peripheral margin of the wound); Major cutaneous abscess: an infection characterized by a collection of pus within the dermis or deeper that is accompanied by redness, edema, and/or induration of a minimum surface area of 75 cm^2 (e.g., the shortest distance of redness, edema, and/or induration extending at least 5 cm from the peripheral margin of the abscess). Cellulitis: a diffuse skin infection characterized by a spreading area of redness, edema, and/or induration of a minimum surface area of 75 cm^2 Note: For subjects with more than one type of eligible lesion/wound or with multiple lesions of the same type, the investigator must clearly identify the lesion to be evaluated for study purposes. The identified lesion must be consistently chosen for assessment (including digital imaging) throughout the study. Incision and drainage (I&D) of the lesion is permitted prior to the first dose of study medication and will be allowed, per protocol, up to 24 hours after the start of the first dose of study medication.
* The subject has at least 1 additional sign or symptom of skin infection: fluctuation, heat/localized warmth, and pain/tenderness.
* The subject has at least 1 systemic marker of infection at the time of screening: Lymphadenopathy (proximal to and within the drainage of the wound); Fever (>=38 degrees Celsius); white blood cells (WBC) elevation (>10000 /cubic millimetre [mm^3] or >10% immature neutrophils regardless of WBC count); C-reactive protein > upper limit of normal (ULN). Note: Systemic markers of infection are not required for subjects >70 years of age or for known or suspected (based on blood glucose levels) diabetics.
* The subject has provided written, dated, informed consent and is willing and able to comply with the study protocol.

Exclusion Criteria:

* The subject is pregnant or nursing.
* The subject has an immune-compromising illness; including known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), organ (including bone marrow) transplant recipients, hematological malignancy, and immunosuppressive therapy, including high-dose corticosteroids (e.g., greater than 40mg prednisone or equivalent per day for greater than two weeks).
* Body mass index (BMI)>= 40.0 kilogram per square meter.
* The subject has a serious underlying disease that could be imminently life-threatening, or is unlikely to survive for the duration of the study period.
* The subject has a medical condition or requires medication that may be aggravated by inhibition of acetylcholinesterase, such as: the subject has poorly controlled asthma or chronic obstructive pulmonary disease at baseline, and, in the opinion, of the investigator is not stable on current therapy; the subject has acute severe pain, uncontrolled with conventional medical management; the subject has active peptic ulcer disease; the subject has parkinson's disease; the subject has myasthenia gravis; the subject has history of seizure disorder requiring medications for control. this does not include a history of childhood febrile seizures; the subject has any evidence of mechanical obstruction of the urinary or digestive tracts.
* The subject has had a diagnosis of C. difficile infection (CDI) within 90 days of screening
* The subject has history of seizure disorder requiring medications for control. This does not include a history of childhood febrile seizures.
* The subject is a chronic abuser of alcohol or illicit substances such that it jeopardizes ability to comply with the protocol
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* The subject has a PR Interval <120 or >220 millisecond (msec)
* Corrected QT interval (QTc) >450msec or QTc >480msec for subjects with bundle branch block. Note: The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread. The QTc should be based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period. It is essential that the same method for calculating QTc that was used at a subjects baseline visit be used for that subject for all subsequent visits.
* The subject has QRS duration <70 or >120 msec.
* The subject has pre-existing grade II atrioventricular block or higher, history of significant vasovagal and/or syncopal episodes, episodes of symptomatic bradycardia.
* The subject has recent acute major blood loss with signs of hemodynamic instability.
* The subject has liver function tests: alanine aminotransferase (ALT) >2x ULN; alkaline phosphatase and bilirubin >=1.5xULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* The subject has a current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Subjects with stable Hepatitis B and/or Hepatitis C will be eligible if they meet the liver function test criteria in criterion (ALT >2 × ULN; alkaline phosphatase and bilirubin ≥1.5 × ULN).

Note: All subjects will be screened for Hepatitis B surface antigen and Hepatitis C ribonucleic acid (RNA), but these results will not be used to determine subject eligibility or subject continuation in the study after enrollment.

* The subject has any skin condition or skin infection listed below: Secondarily infected animal/human bite; Infected burn; Infections of chronic ulcerative lesions (including diabetic foot infections and peripheral vascular disease) that are likely to be polymicrobial in nature, or caused by Gram-negative or anaerobic organisms that are unlikely to have a Gram-positive pathogen as the causative agent, (Note: Subjects with diabetic foot infections or peripheral vascular disease are eligible if they have a qualifying ABSSSI but diabetic foot infections are not eligible lesions for investigation); An underlying skin disease, such as pre-existing eczematous dermatitis, with clinical evidence of secondary infection; Suspected or confirmed osteomyelitis; Suspected or confirmed septic arthritis; Uncomplicated ABSSSI such as simple abscess, impetiginous lesions, superficial cellulitis, furunculosis, carbunculosis, or folliculitis; Infected abdominal wounds unable to be surgically closed; Necrotizing fasciitis, rapidly necrotizing infections, gangrenous processes, or decubitus ulcer; An existing abscess that cannot be drained or a wound requiring significant surgical intervention that cannot be performed within 48 hours of initiation of study treatment; Skin infection known or suspected to be due to fungal, parasitic or viral pathogens; or known or suspected to be due to anaerobic bacterial pathogens or Pseudomonas aeruginosa (including ecthyma gangrenosum), or other Gram negative pathogens as the contributing pathogen; Skin infections complicated by the presence of prosthetic materials that are not to be removed such as central venous catheters, permanent cardiac pacemaker battery packs, or joint replacement prostheses.
* The subject has received treatment with a systemic and/or topical antibacterial within 4 days of study entry; EXCEPT for any of following conditions: The subject received a single dose of a short-acting antibacterial (half-life less than 12 hours) drug prior to the first dose of study treatment; The subject has failed a previous ABSSSI regimen (i.e. at least 48 hours of treatment) and has documented lack of microbiological or clinical response to such therapy. A subject enrolled as a failure of a previous antibacterial treatment regimen must EITHER: Show worsening or lack of improvement or worsening in signs and symptoms of infection, including continued or worsening purulence, erythema with or without induration, fluctuation, heat/localized warmth, and pain/tenderness and/or continued or worsening systemic markers of infection OR show microbiological evidence of failure; The subject recently completed a treatment course with an antibacterial drug for an infection other than ABSSSI and the drug does not have antibacterial activity against bacterial pathogens that cause ABSSSI. (Note: topical antiseptics, chorhexidine, and alcohol and soaps for wound care are permitted). For the purposes of these criteria, the information may be obtained via a verbal interview with the subject or from the subject's medical records; information obtained via a verbal interview must be recorded in the subject's medical record.
* The subject has known or suspected severe impairment of renal function, including a calculated creatinine clearance (as calculated using the Cockroft-Gault method) of less than 30 millilitre per minute; requirement for peritoneal dialysis, hemodialysis, or hemofiltration; or oliguria (less than 20 millilitre urine output per hour over 24 hours).
* The subject has known or suspected chronic neutropenia due to suppression of neutrophil production, or is anticipated to develop neutropenia during the course of the study (ie. new chemotherapy subject), with absolute neutrophil count less than 1000 cells/mm^3 (subjects with neutrophil counts as low as 500 cell/mm^3 are eligible if the reduction is due entirely to the acute infectious process).
* The subject has been previously enrolled in this study, or has previously been treated with GSK2140944.
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2015-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Sylmar, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Miramar, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Hazard, Kentucky
  - GSK Investigational Site, Zachary, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Carriere, Mississippi
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Belleville, New Jersey
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Lima, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Channelview, Texas
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Scangarella-Oman NE, Ingraham KA, Tiffany CA, Tomsho L, Van Horn SF, Mayhew DN, Perry CR, Ashton TC, Dumont EF, Huang J, Brown JR, Miller LA. In Vitro Activity and Microbiological Efficacy of Gepotidacin from a Phase 2, Randomized, Multicenter, Dose-Ranging Study in Patients with Acute Bacterial Skin and Skin Structure Infections. Antimicrob Agents Chemother. 2020 Feb 21;64(3):e01302-19. doi: 10.1128/AAC.01302-19. Print 2020 Feb 21. PMID 31818823
- [Derived] O'Riordan W, Tiffany C, Scangarella-Oman N, Perry C, Hossain M, Ashton T, Dumont E. Efficacy, Safety, and Tolerability of Gepotidacin (GSK2140944) in the Treatment of Patients with Suspected or Confirmed Gram-Positive Acute Bacterial Skin and Skin Structure Infections. Antimicrob Agents Chemother. 2017 May 24;61(6):e02095-16. doi: 10.1128/AAC.02095-16. Print 2017 Jun. PMID 28373199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116704 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 centers in the United States from 24 March 2014 to 22 July 2015.
Pre-assignment Details: A total of 126 participants were randomly assigned to study treatment (all randomized population). A total of 122 participants, who received study treatment, were included in the Modified Intent-to-Treat population (mITT) and safety populations. The mITT population is used in overall study numbers and demographic information.
Groups:
- Gepotidacin 750 mg q12h: Participants received GSK2140944 750 milligrams (mg) intravenous (IV) every 12 hours (q12h; twice daily [BID]) on Day 1 and Day 2. Participants switched to oral GSK2140944 1500 mg q12h (BID) at investigator's discretion or continued to receive GSK2140944 750 mg IV q12h (BID) from Day 3 to Day 10.
- Gepotidacin 1000 mg q12h: Participants received GSK2140944 1000 mg IV q12h (BID) on Day 1 and Day 2. Participants switched to oral GSK2140944 2000 mg q12h (BID) at investigator's discretion or continued to receive GSK2140944 1000 mg IV q12h (BID) from Day 3 to Day 10.
- Gepotidacin 1000 mg q8h: Participants received GSK21409447 1000 mg IV every 8 hours (q8h) three times a day (TID) on Day 1 and Day 2 . Participants switched to oral GSK2140944 2000 mg q12h TID at investigator's discretion or continued to receive GSK2140944 1000 mg IV q8h TID from Day 3 to Day 10.
Period: Overall Study
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Started | 58 | 39 | 25
Completed | 51 | 32 | 24
Not Completed | 7 | 7 | 1
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: mITT population: those participants who received study treatment
Groups:
- Gepotidacin 750 mg q12h: Participants received GSK2140944 750 mg IV every 12 hours (q12h; BID) on Day 1 and Day 2. Participants switched to oral GSK2140944 1500 mg q12h (BID) at investigator's discretion or continued to receive GSK2140944 750 mg IV q12h (BID) from Day 3 to Day 10.
- Gepotidacin 1000 mg q8h: Participants received GSK21409447 1000 mg IV q8h TID on Day 1 and Day 2. Participants switched to oral GSK2140944 2000 mg q12h TID at investigator's discretion or continued to receive GSK2140944 1000 mg IV q8h TID from Day 3 to Day 10.
- Total: Total of all reporting groups
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h | Total
Number analyzed (Participants) | 58 | 39 | 25 | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (11.35) | 44.6 (10.76) | 45.8 (12.64) | 44.7 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 5 | 35
  Male | 40 | 27 | 20 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 2 | 0 | 3
  White | 55 | 36 | 24 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of the Cure Rate as Measured by Clinical Response and Outcome at the Early Efficacy Visit Combined With Withdrawal Rate
Description: Cure rate and withdrawal rate data points was jointly assessed in a composite endpoint for all participants who received at least one dose of GSK2140944. Cure rate was defined as the percentage of participants exhibiting clinical improvement (=>20% reduction in overall lesion area) at the early efficacy visit. Withdrawal rate was defined as the percentage of participants who withdrew from study treatment due to a drug-related adverse event (AE) at any point while on treatment.
Time Frame: Up to Day 3
Population: Modified Intent-to-Treat (MITT) population consisted of all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Participants
  Number Cured | 48 | 28 | 23
  Number Withdrawn | 1 | 0 | 0

2. Secondary Outcome: Number of Participants With Clinical Response and Outcome at Early Efficacy Visit
Description: The assessment was used to determine whether to continue the participant in the study. Clinical response was assessed as either a clinical success or a clinical failure and the clinical outcome was subsequently determined programmatically, based on the clinical response. Clinical success was defined as a reduction in the total surface area of the lesion (as calculated by digital imaging) of >=20% compared to Baseline and no administration of additional antibacterial therapy for the lesion under study. Clinical failure was defined as death of participant; increase or insufficient decrease (i.e., <20%) in the area (as calculated by digital imaging) of the lesion or administration of non-trial antibacterial drug therapy for treatment of the lesion under study before the primary efficacy endpoint assessment. In addition when the participant refused to consent to clinical examination, the clinical outcome was assessed as unable to determine with subsequent response as failure.
Time Frame: Up to Day 3
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Participants
  Clinical Success | 48 | 28 | 23
  Clinical Failure | 7 | 7 | 2
  Unable to Determine | 3 | 4 | 0

3. Secondary Outcome: Number of Participants With Clinical Response and Outcome at the Post Therapy Visit (Day 12-18)
Description: as for outcome 2
Time Frame: Day 12 to Day 18
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Participants
  Clinical Success | 52 | 32 | 21
  Clinical Failure | 1 | 1 | 1
  Unable to Determine | 5 | 6 | 3

4. Secondary Outcome: Number of Participants With Clinical Response and Outcome at the Final Follow up Visit (Day 21-28)
Description: The assessment was used to determine whether to continue the participant in the study. Clinical response was assessed as either a clinical success or a clinical failure and the clinical outcome was subsequently determined programmatically, based on the clinical response. Clinical success was defined as no increase in the total surface area of the lesion (as calculated by digital imaging) compared to post therapy visit and no further administration of antibacterial therapy for the lesion under study. Clinical recurrence was defined as death of participant; increase in the area of the lesion compared to post therapy visit or administration of additional antibacterial therapy for the lesion under study before the efficacy endpoint assessment for participants who were a clinical success at post therapy visit. In addition when the participant refused to consent to clinical examination, the clinical outcome was assessed as unable to determine with subsequent response as failure.
Time Frame: Day 21 to Day 28
Population: MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Participants
  Clinical Success | 50 | 28 | 20
  Clinical Failure | 1 | 1 | 1
  Clinical Recurrence | 2 | 1 | 1
  Unable to Determine | 5 | 9 | 3

5. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Early Efficacy Visit for Staphylococcus Aureus (SA) Pathogen in Lesion Sample
Description: The microbiological outcome was determined by comparing Baseline bacteriology lesion sample, to the culture results at early efficacy visit. The corresponding microbiological response (success or failure) by participant was then assigned. Microbiological eradication or persistence was defined as culture documented elimination or presence of Baseline pathogens from a bacteriology specimen taken at early efficacy visit respectively. Participant was considered to have outcome of presumed microbiological eradication or persistence when the participant was a clinical success or clinical failure and no bacteriological specimen was obtained at early efficacy visit respectively. When the determination of Baseline pathogen microbiological response could not be made, the outcome was considered as unable to determine. The data for SA in lesion sample has been presented.
Time Frame: Up to Day 3
Population: Modified Microbiological ITT consisted of all randomized participants who received at least one dose of study medication and had a Gram-positive pathogens identified from their Baseline bacteriology lesion sample.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 37 | 28 | 11
Number of pathogens
  Microbiological Success, Eradication | 0 | 2 | 0
  Microbiological Success, Presumed Eradication | 24 | 17 | 9
  Microbiological Failure, Persistence | 11 | 3 | 2
  Microbiological Failure, Presumed Persistence | 4 | 6 | 0

6. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Early Efficacy Visit for Methicillin-resistant Staphylococcus Aureus (MRSA) in Lesion Sample
Description: The microbiological outcome was determined by comparing Baseline bacteriology lesion sample, to the culture results at early efficacy visit. The corresponding microbiological response (success or failure) by participant was then assigned. Microbiological eradication or persistence was defined as culture documented elimination or presence of Baseline pathogens from a bacteriology specimen taken at early efficacy visit respectively. Participant was considered to have outcome of presumed microbiological eradication or persistence when the participant was a clinical success or clinical failure and no bacteriological specimen was obtained at early efficacy visit respectively. When the determination of Baseline pathogen microbiological response could not be made, the outcome was considered as unable to determine. The data for MRSA in lesion sample has been presented.
Time Frame: Day 3
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 28 | 20 | 5
Number of pathogens
  Microbiological Success, Eradication | 0 | 2 | 0
  Microbiological Success, Presumed Eradication | 18 | 10 | 4
  Microbiological Failure, Persistence | 7 | 3 | 1
  Microbiological Failure, Presumed Persistence | 4 | 5 | 0

7. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Early Efficacy Visit for Methicillin-susceptible Staphylococcus Aureus (MSSA) in Lesion Sample
Description: The microbiological outcome was determined by comparing Baseline bacteriology lesion sample, to the culture results at early efficacy visit. The corresponding microbiological response (success or failure) by participant was then assigned. Microbiological eradication or persistence was defined as culture documented elimination or presence of Baseline pathogens from a bacteriology specimen taken at early efficacy visit respectively. Participant was considered to have outcome of presumed microbiological eradication or persistence when the participant was a clinical success or clinical failure and no bacteriological specimen was obtained at early efficacy visit respectively. When the determination of Baseline pathogen microbiological response could not be made, the outcome was considered as unable to determine. The data for MSSA in lesion sample has been presented.
Time Frame: Up to Day 3
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 10 | 8 | 6
Number of pathogens
  Microbiological Success, Presumed Eradication | 6 | 7 | 5
  Microbiological Failure, Persistence | 4 | 0 | 1
  Microbiological Failure, Presumed Persistence | 0 | 1 | 0

8. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Early Efficacy Visit for Other Gram-positive Aerobic Pathogens in Lesion Sample
Description: The microbiological outcome was determined by comparing Baseline bacteriology lesion sample, to the culture results at early efficacy visit. The corresponding microbiological response (success or failure) by participant was then assigned. Microbiological eradication or persistence was defined as culture documented elimination or presence of Baseline pathogens from a bacteriology specimen taken at early efficacy visit respectively. Participant was considered to have outcome of presumed microbiological eradication or persistence when the participant was a clinical success or clinical failure and no bacteriological specimen was obtained at early efficacy visit respectively. When the determination of Baseline pathogen microbiological response could not be made, the outcome was considered as unable to determine. The data for other Gram-positive aerobic pathogens in lesion sample has been presented.
Time Frame: Up to Day 3
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 4 | 4 | 3
Number of pathogens
  Microbiological Success, Eradication | 2 | 2 | 0
  Microbiological Success, Presumed Eradication | 0 | 1 | 3
  Microbiological Failure, Presumed Persistence | 1 | 1 | 0
  Microbiological Failure, Unable to Determine | 1 | 0 | 0

9. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Early Efficacy Visit for All Gram-positive Aerobic Pathogens in Lesion Sample
Description: The microbiological outcome was determined by comparing Baseline bacteriology lesion sample, to the culture results at early efficacy visit. The corresponding microbiological response (success or failure) by participant was then assigned. Microbiological eradication or persistence was defined as culture documented elimination or presence of Baseline pathogens from a bacteriology specimen taken at early efficacy visit respectively. Participant was considered to have outcome of presumed microbiological eradication or persistence when the participant was a clinical success or clinical failure and no bacteriological specimen was obtained at early efficacy visit respectively. When the determination of Baseline pathogen microbiological response could not be made, the outcome was considered as unable to determine. The data for all Gram-positive aerobic pathogens in lesion sample has been presented.
Time Frame: Up to Day 3
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 40 | 29 | 13
Number of pathogens
  Microbiological Success, Eradication | 2 | 4 | 0
  Microbiological Success, Presumed Eradication | 24 | 18 | 12
  Microbiological Failure, Persistence | 11 | 3 | 2
  Microbiological Failure, Presumed Persistence | 5 | 7 | 0
  Microbiological Failure, Unable to Determine | 1 | 0 | 0

10. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Early Efficacy Visit for SA, MRSA and All Gram-positive Aerobic Pathogens in Blood Sample
Description: The microbiological outcome was determined by comparing Baseline bacteriology blood culture, to the culture results at early efficacy visit. The corresponding microbiological response (success or failure) by participant was then assigned. Microbiological eradication or persistence was defined as culture documented elimination or presence of Baseline pathogens from a bacteriology specimen taken at early efficacy visit respectively. Participant was considered to have outcome of presumed microbiological eradication or persistence when the participant was a clinical success or clinical failure and no bacteriological specimen was obtained at early efficacy visit respectively. When the determination of Baseline pathogen microbiological response could not be made, the outcome was considered as unable to determine. The data for SA, MRSA and all Gram-positive aerobic pathogens in blood sample has been presented.
Time Frame: Up to Day 3
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h
Number analyzed (Participants) | 2
Number of pathogens
  SA, Microbiological Success, Eradication | 2
  MRSA, Microbiological Success, Eradication | 2
  Aerobic, Microbiological Success, Eradication | 2

11. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Post Therapy Visit for SA Pathogen in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at post therapy visit. Corresponding response (success or failure) was then assigned. Microbiological eradication or persistence was culture documented elimination or presence of Baseline pathogens from a specimen taken at post therapy visit respectively. Presence of pathogens which was presumed to be eradicated at early efficacy visit was microbiological recurrence. Presumed microbiological eradication or persistence was when there was a clinical success or failure and no bacteriological specimen was obtained at post therapy respectively. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at post therapy visit for pathogens presumed eradicated at early efficacy visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for SA in lesion sample has been presented.
Time Frame: Day 12 to Day 18
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 37 | 28 | 11
Number of pathogens
  Microbiological Success, Eradication | 3 | 1 | 0
  Microbiological Success, Presumed Eradication | 32 | 24 | 8
  Microbiological Failure, Presumed Persistence | 3 | 2 | 1
  Microbiological Failure, Presumed Recurrence | 1 | 1 | 2

12. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Post Therapy Visit for MRSA in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at post therapy visit. Corresponding response (success or failure) was then assigned. Microbiological eradication or persistence was culture documented elimination or presence of Baseline pathogens from a specimen taken at post therapy visit respectively. Presence of pathogens which was presumed to be eradicated at early efficacy visit was microbiological recurrence. Presumed microbiological eradication or persistence was when there was a clinical success or failure and no bacteriological specimen was obtained post therapy respectively. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at post therapy visit for pathogens presumed eradicated at early efficacy visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for MRSA in lesion sample has been presented.
Time Frame: Day 12 to Day 18
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 28 | 20 | 5
Number of pathogens
  Microbiological Success, Eradication | 3 | 0 | 0
  Microbiological Success, Presumed Eradication | 22 | 17 | 4
  Microbiological Failure, Presumed Persistence | 3 | 2 | 0
  Microbiological Failure, Presumed Recurrence | 1 | 1 | 1

13. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Post Therapy Visit for MSSA in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at post therapy visit. Corresponding response (success or failure) was then assigned. Microbiological eradication or persistence was culture documented elimination or presence of Baseline pathogens from a specimen taken at post therapy visit respectively. Presence of pathogens which was presumed to be eradicated at early efficacy visit was microbiological recurrence. Presumed microbiological eradication or persistence was when there was a clinical success or failure and no bacteriological specimen was obtained post therapy respectively. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at post therapy visit for pathogens presumed eradicated at early efficacy visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for MSSA in lesion sample has been presented.
Time Frame: Day 12 to Day 18
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 10 | 8 | 6
Number of pathogens
  Microbiological Success, Eradication | 0 | 1 | 0
  Microbiological Success, Presumed Eradication | 10 | 7 | 4
  Microbiological Failure, Presumed Persistence | 0 | 0 | 1
  Microbiological Failure, Presumed Recurrence | 0 | 0 | 1

14. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Post Therapy Visit for Other Gram-positive Aerobic Pathogens in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at post therapy visit. Corresponding response (success or failure) was then assigned. Microbiological eradication or persistence was culture documented elimination or presence of Baseline pathogens from a specimen taken at post therapy visit respectively. Presence of pathogens which was presumed to be eradicated at early efficacy visit was microbiological recurrence. Presumed microbiological eradication or persistence was when there was a clinical success or failure and no bacteriological specimen was obtained post therapy respectively. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at post therapy visit for pathogens presumed eradicated at early efficacy visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine.
Time Frame: Day 12 to Day 18
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 4 | 4 | 3
Number of pathogens
  Microbiological Success, Presumed Eradication | 3 | 3 | 2
  Microbiological Failure, Presumed Persistence | 0 | 1 | 0
  Microbiological Failure, Presumed Recurrence | 1 | 0 | 1

15. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Post Therapy Visit for All Gram-positive Aerobic Pathogens in Lesion Sample
Description: as for outcome 14
Time Frame: Day 12 to Day 18
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 40 | 29 | 13
Number of pathogens
  Microbiological Success, Eradication | 3 | 1 | 0
  Microbiological Success, Presumed Eradication | 35 | 27 | 10
  Microbiological Failure, Presumed Persistence | 3 | 3 | 1
  Microbiological Failure, Presumed Recurrence | 2 | 1 | 3

16. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Post Therapy Visit for SA, MRSA and All Gram-positive Aerobic Pathogens in Blood Sample
Description: as for outcome 14
Time Frame: Day 12 to Day 18
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h
Number analyzed (Participants) | 2
Number of pathogens
  SA, Microbiological Success, Presumed Eradication | 2
  MRSA, Microbiological Success,Presumed Eradication | 2
  Aerobic,MicrobiologicalSuccess,PresumedEradication | 2

17. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Follow up Visit for SA Pathogen in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at final follow up visit. Corresponding response (success or failure) was then assigned. Microbiological eradication was culture documented elimination of Baseline pathogens from a bacteriology specimen taken at final follow up visit. Presumed microbiological eradication was when there was a clinical success and no bacteriological specimen was obtained at final follow up visit. Culture documented presence of Baseline pathogens in a bacteriology specimen taken at final follow up visit was microbiological recurrence. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at final follow up visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for SA pathogen in lesion sample has been presented.
Time Frame: Day 21 to Day 28
Population: Modified Microbiological ITT.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 37 | 28 | 11
Number of pathogens
  Microbiological Success, Eradication | 1 | 0 | 0
  Microbiological Success, Presumed Eradication | 33 | 21 | 8
  Microbiological Failure, Presumed Recurrence | 1 | 4 | 0
  Microbiological Failure, Unable to Determine | 4 | 3 | 3

18. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Follow up Visit for MRSA in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at final follow up visit. Corresponding response (success or failure) was then assigned. Microbiological eradication was culture documented elimination of Baseline pathogens from a bacteriology specimen taken at final follow up visit. Presumed microbiological eradication was when there was a clinical success and no bacteriological specimen was obtained at final follow up visit. Culture documented presence of Baseline pathogens in a bacteriology specimen taken at final follow up visit was microbiological recurrence. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at final follow up visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for MRSA pathogen in lesion sample has been presented.
Time Frame: Day 21 to Day 28
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 28 | 20 | 5
Number of pathogens
  Microbiological Success, Eradication | 1 | 0 | 0
  Microbiological Success, Presumed Eradication | 23 | 14 | 4
  Microbiological Failure, Presumed Recurrence | 1 | 3 | 0
  Microbiological Failure, Unable to Determine | 4 | 3 | 1

19. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Follow up Visit for MSSA in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at final follow up visit. Corresponding response (success or failure) was then assigned. Microbiological eradication was culture documented elimination of Baseline pathogens from a bacteriology specimen taken at final follow up visit. Presumed microbiological eradication was when there was a clinical success and no bacteriological specimen was obtained at final follow up visit. Culture documented presence of Baseline pathogens in a bacteriology specimen taken at final follow up visit was microbiological recurrence. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at final follow up visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for MSSA pathogen in lesion sample has been presented.
Time Frame: Day 21 to Day 28
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 10 | 8 | 6
Number of pathogens
  Microbiological Success, Presumed Eradication | 10 | 7 | 4
  Microbiological Failure, Presumed Recurrence | 0 | 1 | 0
  Microbiological Failure, Unable to Determine | 0 | 0 | 2

20. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Follow up Visit for Other Gram-positive Aerobic Pathogens in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at final follow up visit. Corresponding response (success or failure) was then assigned. Microbiological eradication was culture documented elimination of Baseline pathogens from a bacteriology specimen taken at final follow up visit. Presumed microbiological eradication was when there was a clinical success and no bacteriological specimen was obtained at final follow up visit. Culture documented presence of Baseline pathogens in a bacteriology specimen taken at final follow up visit was microbiological recurrence. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at final follow up visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for other Gram-positive aerobic pathogens in lesion sample has been presented.
Time Frame: Day 21 to Day 28
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 4 | 4 | 3
Number of pathogens
  Microbiological Success, Presumed Eradication | 3 | 2 | 2
  Microbiological Failure, Presumed Recurrence | 0 | 1 | 0
  Microbiological Failure, Unable to Determine | 1 | 1 | 1

21. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Follow up Visit for All Gram-positive Aerobic Pathogens in Lesion Sample
Description: Microbiological outcome was determined by comparing Baseline lesion sample, to culture results at final follow up visit. Corresponding response (success or failure) was then assigned. Microbiological eradication was culture documented elimination of Baseline pathogens from a bacteriology specimen taken at final follow up visit. Presumed microbiological eradication was when there was a clinical success and no bacteriological specimen was obtained at final follow up visit. Culture documented presence of Baseline pathogens in a bacteriology specimen taken at final follow up visit was microbiological recurrence. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at final follow up visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for all Gram-positive aerobic pathogens in lesion sample has been presented.
Time Frame: Day 21 to Day 28
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 40 | 29 | 13
Number of pathogens
  Microbiological Success, Eradication | 1 | 0 | 0
  Microbiological Success, Presumed Eradication | 36 | 23 | 10
  Microbiological Failure, Presumed Recurrence | 1 | 5 | 0
  Microbiological Failure, Unable to Determine | 5 | 4 | 4

22. Secondary Outcome: Number of Pathogens With Microbiological Response and Outcome at Follow up Visit for SA, MRSA and All Gram-positive Aerobic Pathogens in Blood Sample
Description: Microbiological outcome was determined by comparing Baseline blood culture, to culture results at final follow up visit. Corresponding response (success or failure) was then assigned. Microbiological eradication was culture documented elimination of Baseline pathogens from a bacteriology specimen taken at final follow up visit. Presumed microbiological eradication was when there was a clinical success and no bacteriological specimen was obtained at final follow up visit. Culture documented presence of Baseline pathogens in a bacteriology specimen taken at final follow up visit was microbiological recurrence. Presumed microbiological recurrence was when there was a clinical failure and no bacteriological specimen was obtained at final follow up visit. When the determination of Baseline pathogen response could not be made, the outcome was unable to determine. Data for SA, MRSA and all Gram-positive aerobic pathogens in lesion sample has been presented.
Time Frame: Day 21 to Day 28
Population: Modified Microbiological ITT population.
Measure: Number; unit: Number of pathogens
Arm/Group | Gepotidacin 750 mg q12h
Number analyzed (Participants) | 2
Number of pathogens
  SA, Microbiological Success, Presumed Eradication | 2
  MRSA,Microbiological Success,Presumed Eradication | 2
  Aerobic,MicrobiologicalSuccess,PresumedEradication | 2

23. Secondary Outcome: Pharmacokinetic (PK) Parameters (From GSK2140944 Plasma Concentration-time Data): Maximum Observed Concentration (Cmax) on IV Therapy
Description: Samples for assessment of PK parameter Cmax was done on at predose, 1, 2, 2.5, 3, 6, 12 hours post dose on Day 1 to 3. The first occurrence of the Cmax was determined directly from the raw concentration-time data. Data for participants while on IV therapy has been presented.
Time Frame: Predose, 1, 2, 2.5, 3, 6, 12 hours post dose on Day 1 to 3
Population: PK Parameter Population consisted of all participants in the PK concentration population for whom valid and evaluable PK parameters were derived. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 50 | 33 | 24
Nanograms per milliliter | 4590 (42.4) | 6059 (29.8) | 8848 (105.5)

24. Secondary Outcome: PK Parameters (From GSK2140944 Plasma Concentration-time Data): Cmax on Oral Dose Therapy
Description: Samples for assessment of PK parameter Cmax was done at Predose, 1, 2, 3 hours after first orally administered drug and one predose time point anytime from Day 7 to 10. The first occurrence of the Cmax was determined directly from the raw concentration-time data. Data for participants while on oral dose therapy has been presented.
Time Frame: Predose, 1, 2, 3 hours after first orally administered drug and Day 7 to 10 (predose)
Population: PK Parameter Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 51 | 33 | 24
Nanograms per milliliter | 2342 (84.7) | 4329 (67.8) | 3858 (94.1)

25. Secondary Outcome: PK Parameters (From GSK2140944 Plasma Concentration-time Data): Time to Cmax (Tmax) on IV Therapy
Description: Samples for assessment of PK parameter tmax was done at predose, 1, 2, 2.5, 3, 6, 12 hours post dose on Day 1 to 3. The time at which Cmax was observed was determined directly from the raw concentration-time data. Data for participants while on IV therapy has been presented.
Time Frame: Predose, 1, 2, 2.5, 3, 6, 12 hours post dose on Day 1 to 3
Population: PK Parameter Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 50 | 33 | 24
Hours | 1.95 [0.00 to 3.05] | 1.90 [0.90 to 3.00] | 1.93 [0.00 to 3.00]

26. Secondary Outcome: PK Parameters (From GSK2140944 Plasma Concentration-time Data): Tmax on Oral Dose Therapy
Description: Samples for assessment of PK parameter tmax was done at Predose, 1, 2, 3 hours after first orally administered drug and one predose time point anytime from Day 7 to 10. The time at which Cmax was observed was determined directly from the raw concentration-time data. Data for participants while on oral dose therapy has been presented.
Time Frame: Predose, 1, 2, 3 hours after first orally administered drug and Day 7 to 10 (predose)
Population: PK Parameter Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 51 | 33 | 24
Hours | 3.00 [0.95 to 12.00] | 2.92 [1.02 to 12.00] | 2.98 [0.98 to 8.00]

27. Secondary Outcome: PK Parameters (From GSK2140944 Plasma Concentration-time Data): Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Time of the Last Quantifiable Concentration [AUC (0-t)] and AUC Over the Dosing Interval [AUC(0-tau)] on IV Therapy
Description: Samples for assessment of PK parameters AUClast and AUC0-tau was done at predose, 1, 2, 2.5, 3, 6, 12 hours post dose on Day 1 to 3. The AUC 0-t and AUC0-tau was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Data for participants while on IV therapy has been presented.
Time Frame: Predose, 1, 2, 2.5, 3, 6, 12 hours post dose on Day 1 to 3
Population: PK Parameter Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanograms per milliliter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 54 | 36 | 24
Hour nanograms per milliliter
  AUClast: number analyzed (Participants) | 50 | 33 | 24
  AUClast | 15992 (36.7) | 20904 (31.8) | 20851 (64.8)
  AUC0-tau: number analyzed (Participants) | 49 | 33 | 22
  AUC0-tau | 16159 (36.3) | 20815 (31.7) | 21499 (66.9)

28. Secondary Outcome: PK Parameters (From GSK2140944 Plasma Concentration-time Data): AUC (0-t) and AUC(0-tau) on Oral Dose Therapy
Description: Samples for assessment of PK parameters AUClast and AUC0-tau was done at predose, 1, 2, 3 hours after first orally administered drug and one predose time point anytime from Day 7 to 10. The AUC 0-t and AUC0-tau was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Data for participants while on oral dose therapy has been presented.
Time Frame: Predose, 1, 2, 3 hours after first orally administered drug and Day 7 to 10 (predose)
Population: PK Parameter Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanograms per milliliter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 51 | 34 | 25
Hour nanograms per milliliter
  AUClast: number analyzed (Participants) | 51 | 33 | 24
  AUClast | 11965 (101.7) | 19308 (98.8) | 15923 (117.4)
  AUC0-tau: number analyzed (Participants) | 44 | 28 | 22
  AUC0-tau | 14404 (78.2) | 24253 (65.4) | 19300 (77.9)

29. Secondary Outcome: Number of Participants Demonstrating a Decrease in GSK2140944 Susceptibility When Comparing Isolates Recovered From Baseline With Those From Any Time Post-Baseline Skin Specimens
Description: Reduction in susceptibility was defined as a >=4-fold increase in minimum inhibitory concentration (MIC) or >=6 millimeter decrease in zone size between an isolate obtained at Baseline and the same pathogen at subsequent visits.
Time Frame: Up to Day 28
Population: Modified MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 40 | 29 | 13
Participants | 0 | 0 | 0

30. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, medically significant or all events of possible drug-induced liver injury with hyperbilirubinemia.
Time Frame: Up to Day 28
Population: Safety population comprised the same set of participants from MITT population and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Participants
  Any AEs | 41 | 25 | 18
  Any SAEs | 1 | 1 | 0

31. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP was measured with the participant in a supine or semi-supine position, having rested in that position for at least 10 minutes. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: Safety population. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Millimeters of mercury
  SBP, ON IV TREATMENT/DAY 1: number analyzed (Participants) | 58 | 38 | 25
  SBP, ON IV TREATMENT/DAY 1 | -2.9 (15.07) | -1.7 (13.90) | -2.4 (9.43)
  SBP, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 25
  SBP, ON IV TREATMENT/DAY 2 | -4.8 (14.63) | 0.3 (13.55) | -1.9 (9.73)
  SBP, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 44 | 25 | 18
  SBP, ON IV TREATMENT/DAY 3 | -1.7 (14.57) | 1.6 (11.25) | -2.1 (13.88)
  SBP, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 17 | 10 | 2
  SBP, ON IV TREATMENT/DAY 4 | -3.2 (14.25) | -1.2 (17.11) | -22.0 (31.11)
  SBP, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 7 | 0
  SBP, ON IV TREATMENT/DAY 5 | -4.8 (17.90) | -1.6 (31.01) |
  SBP, ON IV TREATMENT/DAY 6: number analyzed (Participants) | 10 | 6 | 0
  SBP, ON IV TREATMENT/DAY 6 | -8.0 (14.60) | -2.7 (14.83) |
  SBP, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 5 | 4 | 0
  SBP, ON IV TREATMENT/DAY 7 | -17.0 (16.57) | 2.3 (32.39) |
  SBP, ON IV TREATMENT/DAY 8: number analyzed (Participants) | 3 | 0 | 0
  SBP, ON IV TREATMENT/DAY 8 | -10.3 (29.87) |  |
  SBP, ON IV TREATMENT/DAY 9: number analyzed (Participants) | 2 | 0 | 0
  SBP, ON IV TREATMENT/DAY 9 | 12.0 (1.41) |  |
  SBP, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  SBP, ON IV TREATMENT/DAY 10 | 6.0 (NA) — Only one participant was analyzed. |  |
  SBP, ORAL - FIRST DAY: number analyzed (Participants) | 53 | 34 | 25
  SBP, ORAL - FIRST DAY | 1.6 (13.36) | 2.3 (13.86) | -3.7 (13.59)
  SBP, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 23
  SBP, ORAL - DAY 7-10 | 2.8 (9.14) | 1.9 (10.55) | -0.9 (17.91)
  SBP, POST THERAPY DAY 12-18: number analyzed (Participants) | 53 | 32 | 22
  SBP, POST THERAPY DAY 12-18 | -0.1 (13.71) | 4.5 (11.33) | 4.1 (11.09)
  SBP, FOLLOW UP DAY 21-28: number analyzed (Participants) | 54 | 30 | 23
  SBP, FOLLOW UP DAY 21-28 | 2.5 (12.87) | 2.1 (12.24) | 1.7 (15.60)
  SBP, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  SBP, POST DOSE DAY 3-10 | -23.0 (NA) — Only one participant was analyzed. |  |
  DBP, ON IV TREATMENT/DAY 1: number analyzed (Participants) | 58 | 38 | 25
  DBP, ON IV TREATMENT/DAY 1 | -3.1 (10.28) | -2.9 (10.97) | -2.3 (9.21)
  DBP, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 25
  DBP, ON IV TREATMENT/DAY 2 | -3.5 (10.84) | -0.9 (9.26) | -2.1 (9.77)
  DBP, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 44 | 25 | 18
  DBP, ON IV TREATMENT/DAY 3 | -4.5 (10.98) | -0.9 (9.93) | -3.5 (14.74)
  DBP, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 17 | 10 | 2
  DBP, ON IV TREATMENT/DAY 4 | -1.9 (12.19) | 0.6 (11.19) | -12.5 (30.41)
  DBP, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 7 | 0
  DBP, ON IV TREATMENT/DAY 5 | -0.9 (13.66) | -2.0 (14.83) |
  DBP, ON IV TREATMENT/DAY 6: number analyzed (Participants) | 10 | 6 | 0
  DBP, ON IV TREATMENT/DAY 6 | -1.4 (11.75) | -9.2 (15.38) |
  DBP, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 5 | 4 | 0
  DBP, ON IV TREATMENT/DAY 7 | -1.6 (23.37) | -13.8 (19.09) |
  DBP, ON IV TREATMENT/DAY 8: number analyzed (Participants) | 3 | 0 | 0
  DBP, ON IV TREATMENT/DAY 8 | -0.3 (18.50) |  |
  DBP, ON IV TREATMENT/DAY 9: number analyzed (Participants) | 2 | 0 | 0
  DBP, ON IV TREATMENT/DAY 9 | 13.0 (21.21) |  |
  DBP, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  DBP, ON IV TREATMENT/DAY 10 | 8.0 (NA) — Only one participant was analyzed. |  |
  DBP, ORAL - FIRST DAY: number analyzed (Participants) | 53 | 34 | 25
  DBP, ORAL - FIRST DAY | 0.0 (11.26) | -1.0 (8.44) | -3.4 (12.84)
  DBP, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 23
  DBP, ORAL - DAY 7-10 | -1.2 (9.12) | 0.4 (8.13) | 0.0 (11.13)
  DBP, POST THERAPY DAY 12-18: number analyzed (Participants) | 53 | 32 | 22
  DBP, POST THERAPY DAY 12-18 | 2.2 (9.18) | 2.3 (8.00) | 3.5 (12.23)
  DBP, FOLLOW UP DAY 21-28: number analyzed (Participants) | 54 | 30 | 23
  DBP, FOLLOW UP DAY 21-28 | 2.3 (11.00) | 0.0 (9.94) | 1.2 (13.44)
  DBP, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  DBP, POST DOSE DAY 3-10 | -5.0 (NA) — Only one participant was analyzed. |  |

32. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured with the participant in a supine or semi-supine position, having rested in that position for at least 10 minutes. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Beats per minute
  ON IV TREATMENT/DAY 1: number analyzed (Participants) | 58 | 38 | 25
  ON IV TREATMENT/DAY 1 | -4.5 (11.38) | -3.8 (10.66) | -2.0 (10.39)
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 25
  ON IV TREATMENT/DAY 2 | -6.3 (14.31) | -1.2 (10.66) | -5.2 (10.78)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 44 | 25 | 18
  ON IV TREATMENT/DAY 3 | -7.5 (14.08) | -6.6 (10.28) | -7.1 (12.62)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 17 | 10 | 2
  ON IV TREATMENT/DAY 4 | -11.3 (18.27) | -5.5 (10.37) | -7.0 (12.73)
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 7 | 0
  ON IV TREATMENT/DAY 5 | -15.1 (22.36) | -9.9 (13.50) |
  ON IV TREATMENT/DAY 6: number analyzed (Participants) | 10 | 6 | 0
  ON IV TREATMENT/DAY 6 | -16.9 (21.60) | -11.0 (10.22) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 5 | 4 | 0
  ON IV TREATMENT/DAY 7 | -28.4 (33.57) | -18.0 (16.75) |
  ON IV TREATMENT/DAY 8: number analyzed (Participants) | 3 | 0 | 0
  ON IV TREATMENT/DAY 8 | -32.3 (15.63) |  |
  ON IV TREATMENT/DAY 9: number analyzed (Participants) | 2 | 0 | 0
  ON IV TREATMENT/DAY 9 | -45.5 (31.82) |  |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | -68.0 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 53 | 34 | 25
  ORAL - FIRST DAY | -6.7 (15.43) | -5.6 (13.47) | -7.0 (11.45)
  ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 23
  ORAL - DAY 7-10 | -1.6 (12.35) | -1.8 (10.53) | -5.7 (15.33)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 53 | 32 | 22
  POST THERAPY DAY 12-18 | -1.6 (15.02) | 2.7 (13.38) | -7.0 (16.34)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 54 | 30 | 25
  FOLLOW UP DAY 21-28 | -1.6 (13.59) | -1.1 (10.09) | -2.5 (17.10)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | -15.0 (NA) — Only one participant was analyzed. |  |

33. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured with the participant in a supine or semi-supine position, having rested in that position for at least 10 minutes. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Breaths per minute
  ON IV TREATMENT/DAY 1: number analyzed (Participants) | 58 | 38 | 25
  ON IV TREATMENT/DAY 1 | -0.4 (2.66) | -0.1 (1.64) | 0.7 (2.90)
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 25
  ON IV TREATMENT/DAY 2 | 0.1 (2.28) | -0.3 (2.37) | -0.5 (1.73)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 44 | 25 | 18
  ON IV TREATMENT/DAY 3 | 0.3 (2.80) | -0.6 (1.58) | -0.3 (2.17)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 17 | 10 | 2
  ON IV TREATMENT/DAY 4 | -0.1 (1.78) | -1.0 (1.94) | -1.0 (1.41)
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 7 | 0
  ON IV TREATMENT/DAY 5 | -0.4 (2.22) | -0.7 (1.25) |
  ON IV TREATMENT/DAY 6: number analyzed (Participants) | 10 | 6 | 0
  ON IV TREATMENT/DAY 6 | -0.1 (2.33) | -0.8 (1.47) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 5 | 4 | 0
  ON IV TREATMENT/DAY 7 | -1.2 (2.68) | -1.0 (1.15) |
  ON IV TREATMENT/DAY 8: number analyzed (Participants) | 3 | 0 | 0
  ON IV TREATMENT/DAY 8 | -1.3 (4.16) |  |
  ON IV TREATMENT/DAY 9: number analyzed (Participants) | 2 | 0 | 0
  ON IV TREATMENT/DAY 9 | -4.0 (2.83) |  |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | -6.0 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 53 | 34 | 25
  ORAL - FIRST DAY | 0.4 (2.33) | 0.3 (1.66) | 0.2 (1.92)
  ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 23
  ORAL - DAY 7-10 | -0.2 (2.39) | -0.1 (2.35) | -0.2 (2.04)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 53 | 32 | 22
  POST THERAPY DAY 12-18 | 0.0 (2.94) | -0.3 (1.97) | -0.4 (2.02)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 54 | 30 | 23
  FOLLOW UP DAY 21-28 | -0.6 (2.81) | -0.3 (2.04) | -0.5 (1.78)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | -2.0 (NA) — Only one participant was analyzed. |  |

34. Secondary Outcome: Change From Baseline in Vital Sign: Body Temperature
Description: Body temperature was measured with the participant in a supine or semi-supine position, having rested in that position for at least 10 minutes. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Celcius
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Celcius
  ON IV TREATMENT/DAY 1: number analyzed (Participants) | 58 | 38 | 25
  ON IV TREATMENT/DAY 1 | -0.126 (0.6632) | -0.053 (0.4114) | -0.172 (0.4208)
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 25
  ON IV TREATMENT/DAY 2 | -0.195 (0.6058) | -0.173 (0.4642) | -0.400 (0.5672)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 44 | 25 | 18
  ON IV TREATMENT/DAY 3 | -0.393 (0.5986) | -0.308 (0.4216) | -0.456 (0.7548)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 17 | 10 | 2
  ON IV TREATMENT/DAY 4 | -0.476 (0.7242) | -0.455 (0.5610) | -0.550 (0.2121)
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 7 | 0
  ON IV TREATMENT/DAY 5 | -0.662 (0.8412) | -0.521 (0.6013) |
  ON IV TREATMENT/DAY 6: number analyzed (Participants) | 10 | 6 | 0
  ON IV TREATMENT/DAY 6 | -1.080 (0.9589) | -0.842 (1.0670) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 5 | 4 | 0
  ON IV TREATMENT/DAY 7 | -1.400 (1.1726) | -0.738 (0.8901) |
  ON IV TREATMENT/DAY 8: number analyzed (Participants) | 3 | 0 | 0
  ON IV TREATMENT/DAY 8 | -0.533 (0.6110) |  |
  ON IV TREATMENT/DAY 9: number analyzed (Participants) | 2 | 0 | 0
  ON IV TREATMENT/DAY 9 | -0.800 (0.7071) |  |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | -1.100 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 53 | 34 | 25
  ORAL - FIRST DAY | -0.398 (0.8149) | -0.304 (0.7005) | -0.608 (0.7593)
  ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 23
  ORAL - DAY 7-10 | -0.498 (0.6496) | -0.468 (0.6417) | -0.635 (0.8483)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 53 | 32 | 22
  POST THERAPY DAY 12-18 | -0.485 (0.7579) | -0.439 (0.6764) | -0.645 (0.9379)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 54 | 30 | 23
  FOLLOW UP DAY 21-28 | -0.441 (0.7579) | -0.375 (0.7255) | -0.604 (0.8891)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | -0.200 (NA) — Only one participant was analyzed. |  |

35. Secondary Outcome: Number of Participants With Maximum Post-Baseline Electrocardiogram (ECG) Readings
Description: The 12-lead ECGs was obtained at Day 1, Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28 for corrected QT, using Fridericia formula (QTcF), corrected QT using Bazett's formula (QTcB) and QRS intervals. The number of participants with maximum post-baseline ECG value exceeding the following limits have been reported: QTcB/QTcF interval > 450 and ≤ 480 millisecond (msec), QTcB/QTcF interval > 480 and ≤ 500 msec, QTcB/QTcF interval > 500 msec, QRS interval < 70 msec and QRS interval > 120 msec.
Time Frame: Up to Day 28
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 38 | 25
Participants
  QTcB, Maximum Post-Baseline, <=450 | 27 | 15 | 9
  QTcB, Maximum Post-Baseline, <=450 and <=480 | 28 | 19 | 11
  QTcB, Maximum Post-Baseline, >480 and <=500 | 3 | 4 | 3
  QTcB, Maximum Post-Baseline, >500 | 0 | 0 | 2
  QTcF, Maximum Post-Baseline, <=450 | 47 | 28 | 17
  QTcF, Maximum Post-Baseline, <=450 and <=480 | 11 | 10 | 8
  QRS, Maximum Post-Baseline, 70 - 120 | 56 | 36 | 23
  QRS, Maximum Post-Baseline, >120 | 2 | 2 | 2

36. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Follicle Stimulating Hormone (FSH) and Gamma Glutamyl Transferase (GGT)
Description: Blood samples for assessment of clinical chemistry parameters of ALT, ALP, AST, FSH and GGT was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
International units per liter
  ALT, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  ALT, ON IV TREATMENT/DAY 2 | -1.9 (5.40) | -1.0 (4.67) | 2.3 (14.57)
  ALT, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  ALT, ON IV TREATMENT/DAY 3 | 1.2 (14.63) | 1.4 (9.71) | 1.2 (6.30)
  ALT, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ALT, ON IV TREATMENT/DAY 4 |  | 14.0 (NA) — Only one participant was analyzed. |
  ALT, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 2 | 6 | 0
  ALT, ON IV TREATMENT/DAY 5 | 9.3 (18.27) | 2.8 (9.89) |
  ALT, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  ALT, ON IV TREATMENT/DAY 7 | 37.5 (19.09) | 18.5 (9.19) |
  ALT, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  ALT, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  ALT, ORAL - FIRST DAY | 3.6 (17.52) | 4.1 (11.58) | 5.7 (11.57)
  ALT, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  ALT, ORAL - DAY 7-10 | 6.6 (15.75) | 7.3 (17.74) | 6.3 (12.60)
  ALT, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  ALT, POST THERAPY DAY 12-18 | 12.8 (35.54) | 8.3 (21.90) | 4.2 (16.02)
  ALT, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 5 | 3
  ALT, FOLLOW UP DAY 21-28 | 36.2 (53.78) | 27.8 (39.03) | 9.3 (4.62)
  ALT, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  ALT, POST DOSE DAY 3-10 | 22.0 (NA) — Only one participant was analyzed. |  |
  ALP, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  ALP, ON IV TREATMENT/DAY 2 | -1.4 (11.52) | -1.3 (12.27) | -4.0 (12.23)
  ALP, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  ALP, ON IV TREATMENT/DAY 3 | 1.8 (18.97) | 5.7 (14.17) | -0.4 (6.17)
  ALP, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ALP, ON IV TREATMENT/DAY 4 |  | 15.0 (NA) — Only one participant was analyzed. |
  ALP, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  ALP, ON IV TREATMENT/DAY 5 | -0.3 (13.01) | 5.0 (11.49) |
  ALP, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  ALP, ON IV TREATMENT/DAY 7 | 3.0 (22.63) | 10.0 (21.21) |
  ALP, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  ALP, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  ALP, ORAL - FIRST DAY | 5.1 (19.30) | 4.0 (17.38) | -0.4 (11.32)
  ALP, ORAL - DAY 7-10: number analyzed (Participants) | 44 | 30 | 21
  ALP, ORAL - DAY 7-10 | 3.8 (13.21) | 2.2 (19.16) | -0.1 (11.17)
  ALP, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  ALP, POST THERAPY DAY 12-18 | -0.8 (15.97) | 0.1 (16.16) | -1.8 (11.72)
  ALP, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 5 | 3
  ALP, FOLLOW UP DAY 21-28 | 4.6 (19.49) | 15.6 (20.84) | -2.0 (3.61)
  ALP, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  ALP, POST DOSE DAY 3-10 | 17.0 (NA) — Only one participant was analyzed. |  |
  AST, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 55 | 35 | 24
  AST, ON IV TREATMENT/DAY 2 | -1.1 (6.58) | 0.7 (7.03) | 2.0 (10.85)
  AST, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  AST, ON IV TREATMENT/DAY 3 | 1.6 (12.47) | 6.2 (22.30) | 6.9 (18.84)
  AST, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  AST, ON IV TREATMENT/DAY 4 |  | 22.0 (NA) — Only one participant was analyzed. |
  AST, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  AST, ON IV TREATMENT/DAY 5 | 7.4 (17.95) | 4.2 (13.01) |
  AST, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 1 | 2 | 0
  AST, ON IV TREATMENT/DAY 7 | 23.0 (NA) — Only one participant was analyzed. | 22.0 (0.00) |
  AST, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  AST, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  AST, ORAL - FIRST DAY | 4.3 (13.34) | 34 (13.52) | 6.3 (17.83)
  AST, ORAL - DAY 7-10: number analyzed (Participants) | 44 | 30 | 21
  AST, ORAL - DAY 7-10 | 6.7 (12.08) | 6.8 (13.93) | 2.3 (17.44)
  AST, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  AST, POST THERAPY DAY 12-18 | 10.9 (18.98) | 9.0 (15.53) | 0.8 (19.05)
  AST, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 5 | 3
  AST, FOLLOW UP DAY 21-28 | 16.2 (22.15) | 22.6 (29.90) | 5.3 (2.52)
  AST, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  AST, POST DOSE DAY 3-10 | 9.0 (NA) — Only one participant was analyzed. |  |
  GGT, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  GGT, ON IV TREATMENT/DAY 2 | -1.5 (7.68) | -1.9 (8.10) | -1.4 (10.15)
  GGT, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  GGT, ON IV TREATMENT/DAY 3 | 1.7 (18.66) | 3.8 (12.23) | 1.9 (5.16)
  GGT, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  GGT, ON IV TREATMENT/DAY 4 |  | -4.0 (NA) — Only one participant was analyzed. |
  GGT, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  GGT, ON IV TREATMENT/DAY 5 | 3.3 (21.70) | -2.5 (5.21) |
  GGT, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  GGT, ON IV TREATMENT/DAY 7 | 25.5 (0.71) | -3.0 (12.73) |
  GGT, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  GGT, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  GGT, ORAL - FIRST DAY | 3.3 (20.16) | 4.5 (16.25) | -1.1 (10.95)
  GGT, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  GGT, ORAL - DAY 7-10 | 3.6 (17.06) | 7.5 (19.89) | -2.2 (14.75)
  GGT, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  GGT, POST THERAPY DAY 12-18 | 3.0 (15.60) | 5.3 (21.08) | -3.9 (16.80)
  GGT, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  GGT, FOLLOW UP DAY 21-28 | 6.0 (13.56) | 64.0 (89.91) | 3.0 (NA) — Only one participant was analyzed.
  GGT, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  GGT, POST DOSE DAY 3-10 | 39.0 (NA) — Only one participant was analyzed. |  |

37. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples for assessment of clinical chemistry parameters of albumin and total protein was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Gram per liter
  Albumin, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Albumin, ON IV TREATMENT/DAY 2 | -2.4 (3.57) | -1.1 (2.93) | -2.9 (3.34)
  Albumin, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Albumin, ON IV TREATMENT/DAY 3 | -1.7 (4.09) | -0.6 (3.52) | -2.0 (3.46)
  Albumin, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Albumin, ON IV TREATMENT/DAY 4 |  | 1.0 (NA) — Only one participant was analyzed. |
  Albumin, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Albumin, ON IV TREATMENT/DAY 5 | -1.1 (4.09) | -1.5 (3.62) |
  Albumin, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Albumin, ON IV TREATMENT/DAY 7 | 4.0 (8.49) | -0.5 (0.71) |
  Albumin, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Albumin, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Albumin, ORAL - FIRST DAY | 0.0 (3.39) | -0.2 (3.37) | -0.9 (2.86)
  Albumin, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Albumin, ORAL - DAY 7-10 | 1.8 (3.58) | 1.4 (3.04) | 1.2 (2.51)
  Albumin, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Albumin, POST THERAPY DAY 12-18 | 2.1 (3.81) | 2.8 (4.41) | 0.8 (3.61)
  Albumin, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Albumin, FOLLOW UP DAY 21-28 | 2.8 (2.36) | 0.3 (2.22) | 0.0 (NA) — Only one participant was analyzed.
  Albumin, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Albumin, POST DOSE DAY 3-10 | -4.0 (NA) — Only one participant was analyzed. |  |
  Protein, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Protein, ON IV TREATMENT/DAY 2 | -3.2 (6.36) | -1.9 (5.86) | -5.2 (6.28)
  Protein, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Protein, ON IV TREATMENT/DAY 3 | -1.6 (7.04) | -0.3 (5.88) | -4.8 (6.59)
  Protein, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Protein, ON IV TREATMENT/DAY 4 |  | 0.0 (NA) — Only one participant was analyzed. |
  Protein, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Protein, ON IV TREATMENT/DAY 5 | -0.5 (8.22) | -2.3 (7.34) |
  Protein, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Protein, ON IV TREATMENT/DAY 7 | 5.5 (13.44) | -1.0 (8.49) |
  Protein, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Protein, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Protein, ORAL - FIRST DAY | 1.4 (5.96) | -0.2 (6.82) | -1.2 (5.05)
  Protein, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Protein, ORAL - DAY 7-10 | 3.1 (6.95) | 2.2 (5.88) | 0.5 (3.59)
  Protein, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Protein, POST THERAPY DAY 12-18 | 2.9 (7.21) | 3.1 (9.14) | -1.1 (5.93)
  Protein, FOLLOW UP DAY 21-28: number analyzed (Participants) | 58 | 4 | 1
  Protein, FOLLOW UP DAY 21-28 | 5.0 (5.29) | 0.8 (5.06) | -7.0 (NA) — Only one participant was analyzed.
  Protein, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Protein, POST DOSE DAY 3-10 | -3.0 (NA) — Only one participant was analyzed. |  |

38. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin and Urate
Description: Blood samples for assessment of clinical chemistry parameters of bilirubin, creatinine, direct bilirubin and urate was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Micromoles per liter
  Bilirubin, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Bilirubin, ON IV TREATMENT/DAY 2 | -1.9 (3.22) | -1.3 (2.87) | -2.4 (3.34)
  Bilirubin, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Bilirubin, ON IV TREATMENT/DAY 3 | -2.8 (4.42) | -1.0 (3.61) | -2.2 (2.73)
  Bilirubin, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Bilirubin, ON IV TREATMENT/DAY 4 |  | -4.0 (NA) — Only one participant was analyzed. |
  Bilirubin, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Bilirubin, ON IV TREATMENT/DAY 5 | -2.8 (4.64) | -4.0 (2.53) |
  Bilirubin, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Bilirubin, ON IV TREATMENT/DAY 7 | 0.0 (0.0) | -4.0 (0.00) |
  Bilirubin, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Bilirubin, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Bilirubin, ORAL - FIRST DAY | -1.9 (3.87) | -1.7 (3.12) | -2.4 (2.69)
  Bilirubin, ORAL - DAY 7-10: number analyzed (Participants) | 44 | 30 | 21
  Bilirubin, ORAL - DAY 7-10 | -0.9 (4.17) | -0.7 (2.49) | -1.7 (2.55)
  Bilirubin, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Bilirubin, POST THERAPY DAY 12-18 | -1.0 (4.35) | -0.5 (3.25) | -1.4 (3.83)
  Bilirubin, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 5 | 3
  Bilirubin, FOLLOW UP DAY 21-28 | 0.0 (8.72) | 0.0 (4.69) | -1.3 (6.11)
  Bilirubin, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Bilirubin, POST DOSE DAY 3-10 | -2.0 (NA) — Only one participant was analyzed. |  |
  Creatinine, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Creatinine, ON IV TREATMENT/DAY 2 | 3.45 (11.885) | -2.33 (19.886) | 0.66 (8.711)
  Creatinine, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Creatinine, ON IV TREATMENT/DAY 3 | 1.30 (10.462) | -5.35 (28.787) | -3.93 (12.123)
  Creatinine, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Creatinine, ON IV TREATMENT/DAY 4 |  | -1.70 (NA) — Only one participant was analyzed. |
  Creatinine, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Creatinine, ON IV TREATMENT/DAY 5 | -0.91 (10.541) | 7.37 (8.704) |
  Creatinine, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Creatinine, ON IV TREATMENT/DAY 7 | 8.40 (10.607) | 6.65 (8.132) |
  Creatinine, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Creatinine, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Creatinine, ORAL - FIRST DAY | 4.22 (11.115) | -3.78 (27.598) | 2.37 (10.268)
  Creatinine, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Creatinine, ORAL - DAY 7-10 | 4.65 (9.930) | 0.72 (30.659) | 4.13 (9.518)
  Creatinine, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Creatinine, POST THERAPY DAY 12-18 | 3.82 (10.641) | 2.93 (26.419) | 2.08 (9.293)
  Creatinine, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Creatinine, FOLLOW UP DAY 21-28 | 9.92 (12.289) | -1.80 (2.846) | 2.70 (NA) — Only one participant was analyzed.
  Creatinine, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Creatinine, POST DOSE DAY 3-10 | -2.70 (NA) — Only one participant was analyzed. |  |
  Direct Bilirubin, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Direct Bilirubin, ON IV TREATMENT/DAY 2 | -0.3 (2.09) | -0.6 (1.79) | -1.1 (2.28)
  Direct Bilirubin, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Direct Bilirubin, ON IV TREATMENT/DAY 3 | -0.2 (2.33) | -0.7 (1.83) | -1.3 (2.24)
  Direct Bilirubin, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Direct Bilirubin, ON IV TREATMENT/DAY 4 |  | -2.0 (NA) — Only one participant was analyzed. |
  Direct Bilirubin, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Direct Bilirubin, ON IV TREATMENT/DAY 5 | -1.0 (1.94) | -0.7 (2.73) |
  Direct Bilirubin, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Direct Bilirubin, ON IV TREATMENT/DAY 7 | -1.0 (1.41) | -3.0 (1.41) |
  Direct Bilirubin, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Direct Bilirubin, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Direct Bilirubin, ORAL - FIRST DAY | -0.4 (2.15) | -0.2 (2.19) | -1.0 (2.08)
  Direct Bilirubin, ORAL - DAY 7-10: number analyzed (Participants) | 44 | 30 | 21
  Direct Bilirubin, ORAL - DAY 7-10 | 0.0 (1.95) | 0.0 (2.10) | -1.0 (2.16)
  Direct Bilirubin, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Direct Bilirubin, POST THERAPY DAY 12-18 | -0.3 (2.02) | 0.0 (1.68) | -1.2 (2.03)
  Direct Bilirubin, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Direct Bilirubin, FOLLOW UP DAY 21-28 | 1.5 (5.00) | 0.5 (1.91) | 0.0 (NA) — Only one participant was analyzed.
  Direct Bilirubin, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Direct Bilirubin, POST DOSE DAY 3-10 | 0.0 (NA) — Only one participant was analyzed. |  |
  Urate, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Urate, ON IV TREATMENT/DAY 2 | 1.2 (44.16) | -11.7 (42.46) | -17.1 (50.43)
  Urate, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Urate, ON IV TREATMENT/DAY 3 | 4.2 (66.33) | 5.7 (52.02) | -14.4 (97.10)
  Urate, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Urate, ON IV TREATMENT/DAY 4 |  | 60.0 (NA) — Only one participant was analyzed. |
  Urate, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Urate, ON IV TREATMENT/DAY 5 | 26.0 (89.47) | 46.7 (50.86) |
  Urate, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Urate, ON IV TREATMENT/DAY 7 | 10.0 (169.71) | 90.0 (28.28) |
  Urate, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Urate, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Urate, ORAL - FIRST DAY | 16.3 (52.46) | 2.9 (67.26) | -1.3 (67.71)
  Urate, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Urate, ORAL - DAY 7-10 | 51.6 (55.31) | 67.0 (69.79) | 55.2 (65.32)
  Urate, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Urate, POST THERAPY DAY 12-18 | 60.8 (73.88) | 49.4 (83.24) | 45.3 (60.31)
  Urate, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Urate, FOLLOW UP DAY 21-28 | 7.5 (80.16) | 10.0 (102.31) | 140.0 (NA) — Only one participant was analyzed.
  Urate, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Urate, POST DOSE DAY 3-10 | 70.0 (NA) — Only one participant was analyzed. |  |

39. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Calcium, Carbon Dioxide, Chloride, Glucose, Magnesium, Potassium, Sodium and Urea
Description: Blood samples for assessment of clinical chemistry parameters of calcium, carbon dioxide, chloride, glucose, magnesium, potassium, sodium and urea was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Millimole per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Millimole per liter
  Calcium, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 55 | 35 | 24
  Calcium, ON IV TREATMENT/DAY 2 | -0.041 (0.1095) | -0.018 (0.1227) | -0.048 (0.1221)
  Calcium, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Calcium, ON IV TREATMENT/DAY 3 | -0.007 (0.1732) | 0.019 (0.1247) | -0.009 (0.1289)
  Calcium, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Calcium, ON IV TREATMENT/DAY 4 |  | -0.180 (NA) — Only one participant was analyzed. |
  Calcium, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Calcium, ON IV TREATMENT/DAY 5 | 0.024 (0.1313) | -0.007 (0.1440) |
  Calcium, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 1 | 2 | 0
  Calcium, ON IV TREATMENT/DAY 7 | 0.080 (NA) — Only one participant was analyzed. | 0.040 (0.2263) |
  Calcium, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Calcium, ORAL - FIRST DAY: number analyzed (Participants) | 50 | 34 | 23
  Calcium, ORAL - FIRST DAY | 0.042 (0.1152) | 0.022 (0.1245) | 0.018 (0.0908)
  Calcium, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Calcium, ORAL - DAY 7-10 | 0.093 (0.1373) | 0.064 (0.1063) | 0.030 (0.1231)
  Calcium, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Calcium, POST THERAPY DAY 12-18 | 0.083 (0.1440) | 0.087 (0.1363) | 0.047 (0.1239)
  Calcium, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 39 | 1
  Calcium, FOLLOW UP DAY 21-28 | 0.090 (0.1685) | 0.060 (0.0673) | 0.060 (NA) — Only one participant was analyzed.
  Calcium, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Calcium, POST DOSE DAY 3-10 | -0.040 (NA) — Only one participant was analyzed. |  |
  Carbon Dioxide, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 55 | 35 | 24
  Carbon Dioxide, ON IV TREATMENT/DAY 2 | -0.5 (2.87) | -0.3 (2.46) | 0.1 (2.49)
  Carbon Dioxide, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Carbon Dioxide, ON IV TREATMENT/DAY 3 | -0.5 (3.34) | -0.6 (2.71) | 0.4 (2.19)
  Carbon Dioxide, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Carbon Dioxide, ON IV TREATMENT/DAY 4 |  | 1.0 (NA) — only one participant was analyzed. |
  Carbon Dioxide, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Carbon Dioxide, ON IV TREATMENT/DAY 5 | 0.1 (4.28) | 0.7 (3.39) |
  Carbon Dioxide, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 1 | 2 | 0
  Carbon Dioxide, ON IV TREATMENT/DAY 7 | 6.0 (NA) — Only one participant was analyzed. | 2.5 (2.12) |
  Carbon Dioxide, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Carbon Dioxide, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Carbon Dioxide, ORAL - FIRST DAY | -0.5 (3.14) | 0.1 (2.55) | -0.4 (2.97)
  Carbon Dioxide, ORAL - DAY 7-10: number analyzed (Participants) | 44 | 30 | 21
  Carbon Dioxide, ORAL - DAY 7-10 | -0.5 (2.43) | 0.4 (2.87) | -0.2 (3.09)
  Carbon Dioxide, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Carbon Dioxide, POST THERAPY DAY 12-18 | -0.3 (2.83) | -0.1 (3.32) | 1.0 (1.73)
  Carbon Dioxide, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Carbon Dioxide, FOLLOW UP DAY 21-28 | -1.5 (3.32) | 2.3 (1.89) | 1.0 (NA) — Only one participant was analyzed.
  Carbon Dioxide, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Carbon Dioxide, POST DOSE DAY 3-10 | -4.0 (NA) — Only one participant was analyzed. |  |
  Chloride, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Chloride, ON IV TREATMENT/DAY 2 | 2.1 (2.32) | 1.3 (2.92) | 2.4 (2.98)
  Chloride, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Chloride, ON IV TREATMENT/DAY 3 | 2.3 (2.92) | 1.4 (2.78) | 2.1 (4.04)
  Chloride, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Chloride, ON IV TREATMENT/DAY 4 |  | -1.0 (NA) — Only one participant was analyzed. |
  Chloride, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Chloride, ON IV TREATMENT/DAY 5 | 2.9 (2.73) | 0.5 (1.05) |
  Chloride, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Chloride, ON IV TREATMENT/DAY 7 | -0.5 (0.71) | 0.5 (0.71) |
  Chloride, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Chloride, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Chloride, ORAL - FIRST DAY | 1.4 (2.52) | 0.4 (2.70) | 1.1 (3.13)
  Chloride, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Chloride, ORAL - DAY 7-10 | 0.8 (3.63) | 0.7 (2.23) | 1.2 (2.93)
  Chloride, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 25
  Chloride, POST THERAPY DAY 12-18 | 1.7 (2.75) | 1.6 (3.21) | 1.8 (2.95)
  Chloride, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Chloride, FOLLOW UP DAY 21-28 | 0.5 (4.93) | -3.0 (2.94) | 3.0 (NA) — Only one participant was analyzed.
  Chloride, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Chloride, POST DOSE DAY 3-10 | 4.0 (NA) — Only one participant was analyzed. |  |
  Glucose, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Glucose, ON IV TREATMENT/DAY 2 | 0.32 (1.973) | -0.31 (2.863) | -0.88 (2.462)
  Glucose, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Glucose, ON IV TREATMENT/DAY 3 | 0.40 (2.144) | 0.48 (3.087) | -0.37 (2.384)
  Glucose, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Glucose, ON IV TREATMENT/DAY 4 |  | 6.60 (NA) — Only one participant was analyzed. |
  Glucose, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Glucose, ON IV TREATMENT/DAY 5 | -0.51 (3.257) | 1.92 (1.723) |
  Glucose, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Glucose, ON IV TREATMENT/DAY 7 | -2.65 (4.313) | 3.70 (2.687) |
  Glucose, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Glucose, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Glucose, ORAL - FIRST DAY | 0.11 (2.115) | 0.13 (2.926) | -0.04 (1.619)
  Glucose, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Glucose, ORAL - DAY 7-10 | 0.14 (1.698) | 1.08 (3.066) | -0.46 (1.741)
  Glucose, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Glucose, POST THERAPY DAY 12-18 | -0.19 (1.774) | 0.34 (2.719) | -0.84 (2.068)
  Glucose, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Glucose, FOLLOW UP DAY 21-28 | -0.38 (1.284) | 1.95 (3.450) | -0.10 (NA) — Only one participant was analyzed.
  Glucose, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Glucose, POST DOSE DAY 3-10 | 0.30 (NA) — Only one participant was analyzed. |  |
  Magnesium, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Magnesium, ON IV TREATMENT/DAY 2 | -0.013 (0.0682) | -0.017 (0.0688) | 0.004 (0.0865)
  Magnesium, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Magnesium, ON IV TREATMENT/DAY 3 | 0.007 (0.0829) | -0.012 (0.0553) | 0.018 (0.0689)
  Magnesium, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Magnesium, ON IV TREATMENT/DAY 4 |  | 0.000 (NA) — Only one participant was analyzed. |
  Magnesium, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Magnesium, ON IV TREATMENT/DAY 5 | 0.044 (0.0532) | -0.040 (0.0738) |
  Magnesium, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Magnesium, ON IV TREATMENT/DAY 7 | 0.140 (0.0000) | -0.080 (0.0283) |
  Magnesium, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Magnesium, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Magnesium, ORAL - FIRST DAY | -0.009 (0.0709) | -0.016 (0.0592) | 0.006 (0.0613)
  Magnesium, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Magnesium, ORAL - DAY 7-10 | 0.006 (0.0810) | -0.007 (0.0708) | 0.021 (0.0659)
  Magnesium, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Magnesium, POST THERAPY DAY 12-18 | -0.005 (0.0864) | 0.006 (0.0870) | -0.008 (0.0737)
  Magnesium, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Magnesium, FOLLOW UP DAY 21-28 | 0.000 (0.1347) | -0.040 (0.0283) | 0.000 (NA) — Only one participant was analyzed.
  Magnesium, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Magnesium, POST DOSE DAY 3-10 | -0.040 (NA) — Only one participant was analyzed. |  |
  Potassium, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 35 | 24
  Potassium, ON IV TREATMENT/DAY 2 | 0.15 (0.398) | 0.07 (0.481) | 0.22 (0.458)
  Potassium, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 32 | 21 | 9
  Potassium, ON IV TREATMENT/DAY 3 | 0.24 (0.353) | 0.11 (0.429) | 0.16 (0.433)
  Potassium, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Potassium, ON IV TREATMENT/DAY 4 |  | -0.10 (NA) — Only one participant was analyzed. |
  Potassium, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Potassium, ON IV TREATMENT/DAY 5 | 0.28 (0.559) | 0.02 (0.183) |
  Potassium, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 0 | 2 | 0
  Potassium, ON IV TREATMENT/DAY 7 |  | 0.55 (0.495) |
  Potassium, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Potassium, ORAL - FIRST DAY: number analyzed (Participants) | 50 | 34 | 23
  Potassium, ORAL - FIRST DAY | 0.36 (0.374) | 0.20 (0.468) | 0.27 (0.365)
  Potassium, ORAL - DAY 7-10: number analyzed (Participants) | 44 | 30 | 21
  Potassium, ORAL - DAY 7-10 | 0.29 (0.483) | 0.06 (0.434) | 0.05 (0.533)
  Potassium, POST THERAPY DAY 12-18: number analyzed (Participants) | 51 | 32 | 19
  Potassium, POST THERAPY DAY 12-18 | 0.28 (0.543) | 0.06 (0.573) | 0.22 (0.487)
  Potassium, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Potassium, FOLLOW UP DAY 21-28 | 1.03 (0.877) | -0.35 (0.998) | 0.60 (NA) — Only one participant was analyzed.
  Potassium, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Potassium, POST DOSE DAY 3-10 | -0.10 (NA) — Only one participant was analyzed. |  |
  Sodium, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Sodium, ON IV TREATMENT/DAY 2 | 1.1 (2.34) | 0.9 (2.67) | 1.6 (1.93)
  Sodium, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Sodium, ON IV TREATMENT/DAY 3 | 1.2 (2.59) | 1.0 (2.65) | 1.4 (4.16)
  Sodium, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Sodium, ON IV TREATMENT/DAY 4 |  | -3.0 (NA) — Only one participant was analyzed. |
  Sodium, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Sodium, ON IV TREATMENT/DAY 5 | 2.8 (2.78) | 1.0 (2.90) |
  Sodium, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Sodium, ON IV TREATMENT/DAY 7 | 2.0 (2.83) | 0.0 (8.49) |
  Sodium, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Sodium, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Sodium, ORAL - FIRST DAY | 1.2 (2.55) | 0.3 (3.05) | 1.2 (2.54)
  Sodium, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Sodium, ORAL - DAY 7-10 | 0.8 (2.44) | 0.5 (2.90) | 1.3 (2.55)
  Sodium, POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  Sodium, POST THERAPY DAY 12-18 | 1.1 (2.53) | 1.4 (2.70) | 1.8 (2.93)
  Sodium, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Sodium, FOLLOW UP DAY 21-28 | -3.0 (2.71) | -2.3 (2.87) | 1.0 (NA) — Only one participant was analyzed.
  Sodium, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Sodium, POST DOSE DAY 3-10 | 5.0 (NA) — Only one participant was analyzed. |  |
  Urea, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  Urea, ON IV TREATMENT/DAY 2 | -0.11 (1.308) | -0.11 (1.189) | -0.58 (1.110)
  Urea, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  Urea, ON IV TREATMENT/DAY 3 | -0.12 (1.484) | -0.24 (1.715) | -0.61 (2.088)
  Urea, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Urea, ON IV TREATMENT/DAY 4 |  | -1.00 (NA) — Only one participant was analyzed. |
  Urea, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  Urea, ON IV TREATMENT/DAY 5 | -0.50 (1.414) | 0.42 (1.320) |
  Urea, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  Urea, ON IV TREATMENT/DAY 7 | 1.00 (2.121) | -0.25 (1.061) |
  Urea, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  Urea, ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  Urea, ORAL - FIRST DAY | -0.13 (1.360) | -0.56 (1.650) | -0.41 (1.379)
  Urea, ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  Urea, ORAL - DAY 7-10 | 0.77 (1.576) | 0.10 (1.945) | 0.29 (1.586)
  Urea, POST THERAPY DAY 12-18: number analyzed (Participants) | 51 | 32 | 19
  Urea, POST THERAPY DAY 12-18 | 0.60 (1.563) | 0.63 (1.437) | -0.03 (1.486)
  Urea, FOLLOW UP DAY 21-28: number analyzed (Participants) | 4 | 4 | 1
  Urea, FOLLOW UP DAY 21-28 | 1.63 (2.016) | 0.25 (1.041) | -1.00 (NA) — Only one participant was analyzed.
  Urea, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Urea, POST DOSE DAY 3-10 | 0.00 (NA) — Only one participant was analyzed. |  |

40. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Creatinine Clearance, Estimated
Description: Blood samples for assessment of clinical chemistry parameter of estimated creatinine clearance was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Milliliter per minute
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Milliliter per minute
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 57 | 35 | 24
  ON IV TREATMENT/DAY 2 | -6.8 (22.65) | -1.8 (17.47) | -1.7 (17.98)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 33 | 21 | 9
  ON IV TREATMENT/DAY 3 | -4.8 (32.17) | 1.7 (30.02) | 3.8 (19.70)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ON IV TREATMENT/DAY 4 |  | 5.0 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 10 | 6 | 0
  ON IV TREATMENT/DAY 5 | -17.4 (59.39) | -14.5 (14.92) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 2 | 2 | 0
  ON IV TREATMENT/DAY 7 | -22.0 (29.70) | -9.5 (13.44) |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 0 | 0 | 0
  ORAL - FIRST DAY: number analyzed (Participants) | 51 | 34 | 23
  ORAL - FIRST DAY | -12.6 (32.53) | -1.1 (31.43) | -6.3 (16.45)
  ORAL - DAY 7-10: number analyzed (Participants) | 45 | 30 | 21
  ORAL - DAY 7-10 | -13.2 (29.04) | -9.7 (36.67) | -8.3 (16.53)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 52 | 32 | 19
  POST THERAPY DAY 12-18 | -8.8 (28.55) | -10.4 (24.61) | -5.6 (12.72)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 3 | 4 | 0
  FOLLOW UP DAY 21-28 | -13.7 (25.54) | 3.8 (5.74) |
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | 6.0 (NA) — Only one participant was analyzed. |  |

41. Secondary Outcome: Estradiol Values at Baseline
Description: Blood samples for assessment of clinical chemistry parameter of estradiol was collected at Baseline (Day 1). No post-baseline values were reported.
Time Frame: Baseline (Day 1)
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomole per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 10 | 4 | 2
Picomole per liter | 229.4 (196.66) | 148.8 (153.58) | 23.5 (23.33)

42. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples for assessment of hematology parameters of basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Giga cells per liter
  Basophils, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Basophils, ON IV TREATMENT/DAY 2 | 0.000 (0.0330) | 0.003 (0.0220) | 0.007 (0.0216)
  Basophils, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 29 | 21 | 9
  Basophils, ON IV TREATMENT/DAY 3 | -0.003 (0.0262) | 0.003 (0.0217) | -0.014 (0.0305)
  Basophils, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Basophils, ON IV TREATMENT/DAY 4 |  | -0.020 (NA) — Only one participant was analyzed. |
  Basophils, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Basophils, ON IV TREATMENT/DAY 5 | 0.008 (0.0212) | 0.007 (0.0437) |
  Basophils, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Basophils, ON IV TREATMENT/DAY 7 | 0.013 (0.0206) | 0.000 (NA) — Only one participant was analyzed. |
  Basophils, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Basophils, ON IV TREATMENT/DAY 10 | -0.020 (NA) — Only one participant was analyzed. |  |
  Basophils, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 22
  Basophils, ORAL - FIRST DAY | 0.000 (0.0310) | 0.000 (0.0185) | -0.004 (0.0171)
  Basophils, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Basophils, ORAL - DAY 7-10 | 0.001 (0.0277) | 0.007 (0.0258) | 0.004 (0.0169)
  Basophils, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Basophils, POST THERAPY DAY 12-18 | 0.005 (0.0304) | 0.001 (0.0217) | 0.001 (0.0190)
  Basophils, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Basophils, FOLLOW UP DAY 21-28 | 0.016 (0.0114) | -0.020 (NA) — Only one participant was analyzed. | -0.007 (0.0404)
  Basophils, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Basophils, POST DOSE DAY 3-10 | 0.040 (NA) — Only one participant was analyzed. |  |
  Eosinophils, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Eosinophils, ON IV TREATMENT/DAY 2 | 0.021 (0.1597) | 0.055 (0.1414) | 0.052 (0.0744)
  Eosinophils, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 29 | 21 | 9
  Eosinophils, ON IV TREATMENT/DAY 3 | 0.010 (0.1405) | 0.024 (0.1474) | 0.016 (0.0995)
  Eosinophils, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Eosinophils, ON IV TREATMENT/DAY 4 |  | 0.250 (NA) — Only one participant was analyzed. |
  Eosinophils, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Eosinophils, ON IV TREATMENT/DAY 5 | 0.026 (0.0826) | 0.025 (0.1245) |
  Eosinophils, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Eosinophils, ON IV TREATMENT/DAY 7 | 0.055 (0.1723) | 0.040 (NA) — Only one participant was analyzed. |
  Eosinophils, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Eosinophils, ON IV TREATMENT/DAY 10 | 0.010 (NA) — Only one participant was analyzed. |  |
  Eosinophils, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 22
  Eosinophils, ORAL - FIRST DAY | 0.013 (0.1443) | 0.051 (0.2001) | 0.027 (0.0927)
  Eosinophils, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Eosinophils, ORAL - DAY 7-10 | 0.014 (0.1492) | 0.001 (0.1391) | 0.052 (0.1066)
  Eosinophils, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Eosinophils, POST THERAPY DAY 12-18 | -0.017 (0.1168) | 0.011 (0.1320) | 0.050 (0.1298)
  Eosinophils, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Eosinophils, FOLLOW UP DAY 21-28 | -0.004 (0.0716) | 0.000 (NA) — Only one participant was analyzed. | 0.060 (0.0436)
  Eosinophils, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Eosinophils, POST DOSE DAY 3-10 | 0.360 (NA) — Only one participant was analyzed. |  |
  Leukocytes, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Leukocytes, ON IV TREATMENT/DAY 2 | -1.39 (2.722) | -1.35 (2.251) | -1.47 (2.086)
  Leukocytes, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 29 | 21 | 9
  Leukocytes, ON IV TREATMENT/DAY 3 | -2.04 (3.091) | -1.80 (2.692) | -2.94 (4.222)
  Leukocytes, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Leukocytes, ON IV TREATMENT/DAY 4 |  | -7.10 (NA) — Only one participant was analyzed. |
  Leukocytes, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Leukocytes, ON IV TREATMENT/DAY 5 | -2.49 (4.376) | -2.57 (1.402) |
  Leukocytes, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Leukocytes, ON IV TREATMENT/DAY 7 | -4.55 (5.108) | -2.90 (NA) — Only one participant was analyzed. |
  Leukocytes, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Leukocytes, ON IV TREATMENT/DAY 10 | -11.20 (NA) — Only one participant was analyzed. |  |
  Leukocytes, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 22
  Leukocytes, ORAL - FIRST DAY | -1.31 (2.959) | -2.32 (2.527) | -1.69 (2.641)
  Leukocytes, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Leukocytes, ORAL - DAY 7-10 | -1.08 (2.482) | -1.91 (2.299) | -1.67 (2.637)
  Leukocytes, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Leukocytes, POST THERAPY DAY 12-18 | -2.15 (3.053) | -2.20 (2.464) | -2.25 (3.152)
  Leukocytes, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Leukocytes, FOLLOW UP DAY 21-28 | -2.06 (2.428) | -5.70 (NA) — Only one participant was analyzed. | -3.23 (5.877)
  Leukocytes, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Leukocytes, POST DOSE DAY 3-10 | -12.60 (NA) — Only one participant was analyzed. |  |
  Lymphocytes, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Lymphocytes, ON IV TREATMENT/DAY 2 | 0.019 (0.6137) | 0.009 (0.5047) | 0.358 (0.7229)
  Lymphocytes, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 29 | 21 | 9
  Lymphocytes, ON IV TREATMENT/DAY 3 | 0.263 (0.5574) | 0.094 (0.3504) | 0.129 (0.5742)
  Lymphocytes, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Lymphocytes, ON IV TREATMENT/DAY 4 |  | 0.790 (NA) — Only one participant was analyzed. |
  Lymphocytes, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Lymphocytes, ON IV TREATMENT/DAY 5 | 0.288 (0.6918) | 0.075 (0.5417) |
  Lymphocytes, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Lymphocytes, ON IV TREATMENT/DAY 7 | 0.705 (0.5291) | 0.200 (NA) — Only one participant was analyzed. |
  Lymphocytes, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Lymphocytes, ON IV TREATMENT/DAY 10 | 1.230 (NA) — Only one participant was analyzed. |  |
  Lymphocytes, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 22
  Lymphocytes, ORAL - FIRST DAY | 0.002 (0.6844) | -0.050 (0.7343) | 0.247 (0.8342)
  Lymphocytes, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Lymphocytes, ORAL - DAY 7-10 | 0.222 (0.6592) | 0.204 (0.7131) | 0.284 (0.6655)
  Lymphocytes, POST-THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Lymphocytes, POST-THERAPY DAY 12-18 | 0.179 (0.7122) | 0.028 (0.6588) | 0.184 (0.5295)
  Lymphocytes, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Lymphocytes, FOLLOW UP DAY 21-28 | 0.326 (0.3564) | -0.020 (NA) — Only one participant was analyzed. | 0.097 (0.2743)
  Lymphocytes, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Lymphocytes, POST DOSE DAY 3-10 | 0.850 (NA) — Only one participant was analyzed. |  |
  Monocytes, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Monocytes, ON IV TREATMENT/DAY 2 | -0.054 (0.1938) | -0.030 (0.2160) | -0.011 (0.2524)
  Monocytes, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 29 | 21 | 9
  Monocytes, ON IV TREATMENT/DAY 3 | -0.002 (0.2326) | -0.133 (0.2330) | -0.219 (0.5008)
  Monocytes, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Monocytes, ON IV TREATMENT/DAY 4 |  | -0.280 (NA) — Only one participant was analyzed. |
  Monocytes, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Monocytes, ON IV TREATMENT/DAY 5 | -0.114 (0.2056) | -0.243 (0.2448) |
  Monocytes, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Monocytes, ON IV TREATMENT/DAY 7 | 0.022 (0.3231) | -0.170 (NA) — Only one participant was analyzed. |
  Monocytes, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Monocytes, ON IV TREATMENT/DAY 10 | -0.240 (NA) — Only one participant was analyzed. |  |
  Monocytes, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 22
  Monocytes, ORAL - FIRST DAY | -0.076 (0.2069) | -0.099 (0.2379) | -0.154 (0.2919)
  Monocytes, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Monocytes, ORAL - DAY 7-10 | -0.014 (0.2030) | -0.067 (0.1690) | -0.070 (0.3348)
  Monocytes, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Monocytes, POST THERAPY DAY 12-18 | -0.077 (0.1442) | -0.130 (0.2240) | -0.133 (0.3065)
  Monocytes, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Monocytes, FOLLOW UP DAY 21-28 | 0.018 (0.2969) | 0.050 (NA) — Only one participant was analyzed. | -0.347 (0.7050)
  Monocytes, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Monocytes, POST DOSE DAY 3-10 | 0.280 (NA) — Only one participant was analyzed. |  |
  Neutrophils, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Neutrophils, ON IV TREATMENT/DAY 2 | -1.373 (2.7464) | -1.395 (2.4280) | -1.873 (2.0729)
  Neutrophils, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 29 | 21 | 9
  Neutrophils, ON IV TREATMENT/DAY 3 | -2.324 (3.2252) | -1.789 (2.6403) | -2.854 (3.6332)
  Neutrophils, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Neutrophils, ON IV TREATMENT/DAY 4 |  | -7.880 (NA) — Only one participant was analyzed. |
  Neutrophils, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Neutrophils, ON IV TREATMENT/DAY 5 | -2.712 (4.5024) | -2.445 (0.9370) |
  Neutrophils, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Neutrophils, ON IV TREATMENT/DAY 7 | -5.403 (5.1790) | -2.910 (NA) — Only one participant was analyzed. |
  Neutrophils, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Neutrophils, ON IV TREATMENT/DAY 10 | -12.250 (NA) — Only one participant was analyzed. |  |
  Neutrophils, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 22
  Neutrophils, ORAL - FIRST DAY | -1.244 (3.0855) | -2.229 (2.6921) | -1.802 (2.5066)
  Neutrophils, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Neutrophils, ORAL - DAY 7-10 | -1.363 (2.4532) | -2.068 (2.3963) | -1.930 (2.7752)
  Neutrophils, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Neutrophils, POST THERAPY DAY 12-18 | -2.243 (3.2754) | -2.111 (2.6465) | -2.346 (3.0470)
  Neutrophils, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Neutrophils, FOLLOW UP DAY 21-28 | -2.436 (2.5072) | -5.770 (NA) — Only one participant was analyzed. | -3.007 (5.4347)
  Neutrophils, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Neutrophils, POST DOSE DAY 3-10 | -14.050 (NA) — Only one participant was analyzed. |  |
  Platelets, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 28 | 21
  Platelets, ON IV TREATMENT/DAY 2 | 5.6 (37.64) | 6.3 (41.11) | -6.7 (57.38)
  Platelets, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 20 | 8
  Platelets, ON IV TREATMENT/DAY 3 | 5.8 (44.94) | 3.1 (41.89) | -0.6 (19.64)
  Platelets, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Platelets, ON IV TREATMENT/DAY 4 |  | -30.0 (NA) — only one participant was analyzed. |
  Platelets, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 12 | 6 | 0
  Platelets, ON IV TREATMENT/DAY 5 | 43.7 (78.78) | 21.3 (33.02) |
  Platelets, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Platelets, ON IV TREATMENT/DAY 7 | 77.8 (107.48) | -9.0 (NA) — Only one participant was analyzed. |
  Platelets, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Platelets, ON IV TREATMENT/DAY 10 | 159.0 (NA) — Only one participant was analyzed. |  |
  Platelets, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 28 | 21
  Platelets, ORAL - FIRST DAY | 44.0 (74.12) | 0.1 (73.36) | 11.6 (52.46)
  Platelets, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 28 | 20
  Platelets, ORAL - DAY 7-10 | 22.7 (55.11) | 33.9 (95.63) | 22.0 (63.18)
  Platelets, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 29 | 18
  Platelets, POST THERAPY DAY 12-18 | 17.5 (76.72) | 2.9 (88.15) | 0.6 (56.26)
  Platelets, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Platelets, FOLLOW UP DAY 21-28 | 21.0 (26.44) | -92.0 (NA) — Only one participant was analyzed. | -23.3 (62.93)
  Platelets, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Platelets, POST DOSE DAY 3-10 | 148.0 (NA) — Only one participant was analyzed. |  |

43. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocyte Mean Corpuscular Hemoglobin Concentration (EMCHC) and Hemoglobin
Description: Blood samples for assessment of hematology parameters of EMCHC and hemoglobin was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Gram per liter
  EMCHC, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  EMCHC, ON IV TREATMENT/DAY 2 | 1.2 (6.08) | 2.0 (6.90) | 0.1 (6.94)
  EMCHC, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 21 | 9
  EMCHC, ON IV TREATMENT/DAY 3 | -0.4 (6.64) | 2.9 (7.67) | 2.9 (7.90)
  EMCHC, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  EMCHC, ON IV TREATMENT/DAY 4 |  | 0.0 (NA) — Only one participant was analyzed. |
  EMCHC, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  EMCHC, ON IV TREATMENT/DAY 5 | -4.3 (7.51) | 5.8 (10.85) |
  EMCHC, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  EMCHC, ON IV TREATMENT/DAY 7 | 2.8 (9.60) | 6.0 (NA) — Only one participant was analyzed. |
  EMCHC, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  EMCHC, ON IV TREATMENT/DAY 10 | -6.0 (NA) — Only one participant was analyzed. |  |
  EMCHC, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 23
  EMCHC, ORAL - FIRST DAY | 1.2 (8.08) | 0.9 (8.23) | 1.1 (6.13)
  EMCHC, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  EMCHC, ORAL - DAY 7-10 | 2.8 (5.55) | 2.1 (7.06) | 2.1 (8.46)
  EMCHC, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  EMCHC, POST THERAPY DAY 12-18 | 1.6 (6.49) | 2.1 (6.83) | 0.6 (7.93)
  EMCHC, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  EMCHC, FOLLOW UP DAY 21-28 | 5.6 (10.81) | 0.0 (NA) — Only one participant was analyzed. | 8.3 (13.32)
  EMCHC, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  EMCHC, POST DOSE DAY 3-10 | 21.0 (NA) — Only one participant was analyzed. |  |
  Hemoglobin, ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  Hemoglobin, ON IV TREATMENT/DAY 2 | -3.0 (9.04) | -1.2 (9.10) | -4.0 (8.79)
  Hemoglobin, ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 21 | 9
  Hemoglobin, ON IV TREATMENT/DAY 3 | -2.2 (10.95) | -2.2 (11.13) | -1.6 (8.22)
  Hemoglobin, ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  Hemoglobin, ON IV TREATMENT/DAY 4 |  | -8.0 (NA) — Only one participant was analyzed. |
  Hemoglobin, ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  Hemoglobin, ON IV TREATMENT/DAY 5 | -4.7 (10.27) | -8.0 (13.93) |
  Hemoglobin, ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  Hemoglobin, ON IV TREATMENT/DAY 7 | -9.8 (7.80) | 3.0 (NA) — Only one participant was analyzed. |
  Hemoglobin, ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  Hemoglobin, ON IV TREATMENT/DAY 10 | -24.0 (NA) — Only one participant was analyzed. |  |
  Hemoglobin, ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 23
  Hemoglobin, ORAL - FIRST DAY | 4.2 (9.42) | -0.9 (12.20) | -1.0 (8.20)
  Hemoglobin, ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  Hemoglobin, ORAL - DAY 7-10 | 3.9 (11.18) | 1.8 (9.74) | -0.6 (7.45)
  Hemoglobin, POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  Hemoglobin, POST THERAPY DAY 12-18 | 3.8 (10.18) | 2.2 (9.02) | -0.1 (10.85)
  Hemoglobin, FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  Hemoglobin, FOLLOW UP DAY 21-28 | 8.4 (5.50) | -7.0 (NA) — Only one participant was analyzed. | 3.0 (15.87)
  Hemoglobin, POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  Hemoglobin, POST DOSE DAY 3-10 | -1.0 (NA) — Only one participant was analyzed. |  |

44. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocyte Mean Corpuscular Hemoglobin (EMCH)
Description: Blood samples for assessment of hematology parameter of EMCH was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Picograms
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  ON IV TREATMENT/DAY 2 | 0.11 (0.413) | 0.04 (0.386) | -0.07 (0.354)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 21 | 9
  ON IV TREATMENT/DAY 3 | 0.00 (0.278) | 0.05 (0.495) | -0.03 (0.374)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ON IV TREATMENT/DAY 4 |  | -0.40 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  ON IV TREATMENT/DAY 5 | -0.19 (0.325) | 0.12 (0.319) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  ON IV TREATMENT/DAY 7 | 0.30 (0.294) | 0.20 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | -0.20 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 23
  ORAL - FIRST DAY | 0.08 (0.408) | -0.01 (0.389) | -0.14 (0.333)
  ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  ORAL - DAY 7-10 | 0.01 (0.290) | -0.03 (0.390) | -0.06 (0.438)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  POST THERAPY DAY 12-18 | -0.04 (0.389) | 0.01 (0.366) | -0.08 (0.709)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 25
  FOLLOW UP DAY 21-28 | 0.06 (0.483) | -0.40 (NA) — Only one participant was analyzed. | 1.20 (1.735)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | 0.10 (NA) — Only one participant was analyzed. |  |

45. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocyte Mean Corpuscular Volume (EMCV)
Description: Blood samples for assessment of hematology parameter of EMCV was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Femtoliter
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  ON IV TREATMENT/DAY 2 | 0.0 (1.73) | -0.4 (1.56) | -0.1 (1.90)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 21 | 9
  ON IV TREATMENT/DAY 3 | 0.0 (1.61) | -0.6 (1.63) | -0.9 (1.96)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ON IV TREATMENT/DAY 4 |  | -2.0 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  ON IV TREATMENT/DAY 5 | 0.7 (2.06) | -1.0 (2.68) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  ON IV TREATMENT/DAY 7 | 0.0 (3.65) | -1.0 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | 1.0 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 23
  ORAL - FIRST DAY | 0.0 (1.96) | -0.3 (2.11) | -0.7 (1.66)
  ORAL - DAY 7-10: number analyzed (Participants) | 43 | 31 | 21
  ORAL - DAY 7-10 | -0.8 (1.52) | -0.6 (1.50) | -0.9 (1.77)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 39 | 19
  POST THERAPY DAY 12-18 | -0.6 (1.76) | -0.5 (1.59) | -0.5 (1.68)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  FOLLOW UP DAY 21-28 | -1.6 (1.82) | -2.0 (NA) — Only one participant was analyzed. | 2.3 (3.21)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | -7.0 (NA) — Only one participant was analyzed. |  |

46. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes
Description: Blood samples for assessment of hematology parameter of erythrocyte was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Trillion cells per liter
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  ON IV TREATMENT/DAY 2 | -0.14 (0.332) | -0.04 (0.340) | -0.12 (0.345)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 21 | 9
  ON IV TREATMENT/DAY 3 | -0.09 (0.430) | -0.06 (0.430) | -0.07 (0.320)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ON IV TREATMENT/DAY 4 |  | -0.30 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 39 | 0
  ON IV TREATMENT/DAY 5 | -0.14 (0.373) | -0.28 (0.475) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  ON IV TREATMENT/DAY 7 | -0.35 (0.238) | 0.10 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | -0.80 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 23
  ORAL - FIRST DAY | 0.12 (0.362) | -0.01 (0.420) | -0.01 (0.317)
  ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  ORAL - DAY 7-10 | 0.12 (0.400) | 0.07 (0.383) | -0.01 (0.284)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  POST THERAPY DAY 12-18 | 0.13 (0.360) | 0.07 (0.346) | 0.02 (0.416)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  FOLLOW UP DAY 21-28 | 0.26 (0.182) | -0.20 (NA) — Only one participant was analyzed. | -0.03 (0.351)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | 0.00 (NA) — Only one participant was analyzed. |  |

47. Secondary Outcome: Change From Baseline in Hematology Parameters: Hematocrit
Description: Blood samples for assessment of hematology parameter of hematocrit was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28. Baseline was defined at Day 1. Change from Baseline was calculated by subtracting the post-Baseline value from Baseline value.
Time Frame: Baseline (Day 1) up to Day 28
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Ratio
  ON IV TREATMENT/DAY 2: number analyzed (Participants) | 54 | 30 | 23
  ON IV TREATMENT/DAY 2 | -0.0111 (0.03004) | -0.0065 (0.03316) | -0.0125 (0.03152)
  ON IV TREATMENT/DAY 3: number analyzed (Participants) | 30 | 21 | 9
  ON IV TREATMENT/DAY 3 | -0.0066 (0.03683) | -0.0099 (0.03922) | -0.0073 (0.02536)
  ON IV TREATMENT/DAY 4: number analyzed (Participants) | 0 | 1 | 0
  ON IV TREATMENT/DAY 4 |  | -0.0260 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 5: number analyzed (Participants) | 13 | 6 | 0
  ON IV TREATMENT/DAY 5 | -0.0101 (0.03166) | -0.0322 (0.04462) |
  ON IV TREATMENT/DAY 7: number analyzed (Participants) | 4 | 1 | 0
  ON IV TREATMENT/DAY 7 | -0.0353 (0.01873) | 0.0020 (NA) — Only one participant was analyzed. |
  ON IV TREATMENT/DAY 10: number analyzed (Participants) | 1 | 0 | 0
  ON IV TREATMENT/DAY 10 | -0.0690 (NA) — Only one participant was analyzed. |  |
  ORAL - FIRST DAY: number analyzed (Participants) | 48 | 31 | 23
  ORAL - FIRST DAY | 0.0112 (0.03422) | -0.0041 (0.04091) | -0.0043 (0.02854)
  ORAL - DAY 7-10: number analyzed (Participants) | 43 | 29 | 21
  ORAL - DAY 7-10 | 0.0080 (0.03674) | 0.0027 (0.03459) | -0.0040 (0.02840)
  POST THERAPY DAY 12-18: number analyzed (Participants) | 50 | 31 | 19
  POST THERAPY DAY 12-18 | 0.0100 (0.03340) | 0.0039 (0.02846) | -0.0006 (0.04085)
  FOLLOW UP DAY 21-28: number analyzed (Participants) | 5 | 1 | 3
  FOLLOW UP DAY 21-28 | 0.0178 (0.01699) | -0.0220 (NA) — Only one participant was analyzed. | 0.0033 (0.03988)
  POST DOSE DAY 3-10: number analyzed (Participants) | 1 | 0 | 0
  POST DOSE DAY 3-10 | -0.0320 (NA) — Only one participant was analyzed. |  |

48. Secondary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results
Description: Samples for urinalysis assessment was collected at Baseline (Day 1), Day 2, Day 7 to 10, Day 12 to 21 and Day 21 to Day 28 for Glucose, Ketones, Occult Blood, Protein and pH. Participants with abnormal urinalysis result was reported.
Time Frame: Up to day 28
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
Number analyzed (Participants) | 58 | 39 | 25
Participants
  Glucose, BASELINE/DAY 1, Trace: number analyzed (Participants) | 54 | 37 | 24
  Glucose, BASELINE/DAY 1, Trace | 1 | 2 | 1
  Glucose, BASELINE/DAY 1, 1+: number analyzed (Participants) | 54 | 37 | 24
  Glucose, BASELINE/DAY 1, 1+ | 1 | 1 | 1
  Glucose, BASELINE/DAY 1, 3+: number analyzed (Participants) | 54 | 37 | 24
  Glucose, BASELINE/DAY 1, 3+ | 1 | 2 | 1
  Glucose, ON IV TREATMENT/DAY 2, Trace: number analyzed (Participants) | 58 | 31 | 23
  Glucose, ON IV TREATMENT/DAY 2, Trace | 1 | 0 | 0
  Glucose, ON IV TREATMENT/DAY 2, 1+: number analyzed (Participants) | 58 | 31 | 23
  Glucose, ON IV TREATMENT/DAY 2, 1+ | 0 | 0 | 2
  Glucose, ON IV TREATMENT/DAY 2, 3+: number analyzed (Participants) | 58 | 31 | 23
  Glucose, ON IV TREATMENT/DAY 2, 3+ | 3 | 2 | 1
  Glucose, ON IV TREATMENT/DAY 3, 2+: number analyzed (Participants) | 32 | 20 | 9
  Glucose, ON IV TREATMENT/DAY 3, 2+ | 1 | 1 | 0
  Glucose, ON IV TREATMENT/DAY 3, 3+: number analyzed (Participants) | 32 | 20 | 9
  Glucose, ON IV TREATMENT/DAY 3, 3+ | 1 | 1 | 0
  Glucose, ON IV TREATMENT/DAY 5, 2+: number analyzed (Participants) | 13 | 6 | 0
  Glucose, ON IV TREATMENT/DAY 5, 2+ | 1 | 0 |
  Glucose, ON IV TREATMENT/DAY 7, 2+: number analyzed (Participants) | 4 | 1 | 0
  Glucose, ON IV TREATMENT/DAY 7, 2+ | 1 | 0 |
  Glucose, ORAL - FIRST DAY, Trace: number analyzed (Participants) | 51 | 31 | 22
  Glucose, ORAL - FIRST DAY, Trace | 0 | 1 | 0
  Glucose, ORAL - FIRST DAY, 1+: number analyzed (Participants) | 51 | 31 | 22
  Glucose, ORAL - FIRST DAY, 1+ | 1 | 0 | 0
  Glucose, ORAL - FIRST DAY, 3+: number analyzed (Participants) | 51 | 31 | 22
  Glucose, ORAL - FIRST DAY, 3+ | 1 | 2 | 0
  Glucose, ORAL - DAY 7-10, Trace: number analyzed (Participants) | 45 | 30 | 22
  Glucose, ORAL - DAY 7-10, Trace | 1 | 0 | 0
  Glucose, ORAL - DAY 7-10, 1+: number analyzed (Participants) | 45 | 30 | 22
  Glucose, ORAL - DAY 7-10, 1+ | 0 | 1 | 0
  Glucose, ORAL - DAY 7-10, 2+: number analyzed (Participants) | 45 | 30 | 22
  Glucose, ORAL - DAY 7-10, 2+ | 0 | 1 | 0
  Glucose, ORAL - DAY 7-10, 3+: number analyzed (Participants) | 42 | 30 | 22
  Glucose, ORAL - DAY 7-10, 3+ | 0 | 2 | 0
  Glucose, POST THERAPY DAY 12-18, Trace: number analyzed (Participants) | 53 | 32 | 22
  Glucose, POST THERAPY DAY 12-18, Trace | 3 | 0 | 0
  Glucose, POST THERAPY DAY 12-18, 1+: number analyzed (Participants) | 53 | 32 | 22
  Glucose, POST THERAPY DAY 12-18, 1+ | 0 | 1 | 0
  Glucose, POST THERAPY DAY 12-18, 3+: number analyzed (Participants) | 53 | 32 | 22
  Glucose, POST THERAPY DAY 12-18, 3+ | 0 | 3 | 0
  Ketones, BASELINE/DAY 1, Trace: number analyzed (Participants) | 54 | 37 | 24
  Ketones, BASELINE/DAY 1, Trace | 8 | 3 | 6
  Ketones, BASELINE/DAY 1, 1+: number analyzed (Participants) | 54 | 37 | 24
  Ketones, BASELINE/DAY 1, 1+ | 1 | 1 | 0
  Ketones, BASELINE/DAY 1, 3+: number analyzed (Participants) | 54 | 37 | 24
  Ketones, BASELINE/DAY 1, 3+ | 0 | 2 | 0
  Ketones, ON IV TREATMENT/DAY 2, Trace: number analyzed (Participants) | 58 | 31 | 23
  Ketones, ON IV TREATMENT/DAY 2, Trace | 4 | 3 | 1
  Ketones, ON IV TREATMENT/DAY 2, 1+: number analyzed (Participants) | 58 | 31 | 23
  Ketones, ON IV TREATMENT/DAY 2, 1+ | 2 | 1 | 0
  Ketones, ON IV TREATMENT/DAY 2, 3+: number analyzed (Participants) | 58 | 31 | 23
  Ketones, ON IV TREATMENT/DAY 2, 3+ | 0 | 0 | 1
  Ketones, ON IV TREATMENT/DAY 3, Trace: number analyzed (Participants) | 32 | 20 | 9
  Ketones, ON IV TREATMENT/DAY 3, Trace | 5 | 0 | 2
  Ketones, ORAL - FIRST DAY, Trace: number analyzed (Participants) | 51 | 31 | 22
  Ketones, ORAL - FIRST DAY, Trace | 3 | 1 | 2
  Ketones, ORAL - FIRST DAY, 2+: number analyzed (Participants) | 51 | 31 | 22
  Ketones, ORAL - FIRST DAY, 2+ | 1 | 0 | 0
  Ketones, ORAL - DAY 7-10, Trace: number analyzed (Participants) | 45 | 30 | 22
  Ketones, ORAL - DAY 7-10, Trace | 6 | 3 | 3
  Ketones, POST THERAPY DAY 12-18, Trace: number analyzed (Participants) | 53 | 32 | 22
  Ketones, POST THERAPY DAY 12-18, Trace | 8 | 6 | 2
  Occult Blood, BASELINE/DAY 1, Trace: number analyzed (Participants) | 54 | 37 | 24
  Occult Blood, BASELINE/DAY 1, Trace | 3 | 1 | 1
  Occult Blood, BASELINE/DAY 1, 1+: number analyzed (Participants) | 54 | 37 | 24
  Occult Blood, BASELINE/DAY 1, 1+ | 4 | 0 | 1
  Occult Blood, BASELINE/DAY 1, 2+: number analyzed (Participants) | 54 | 37 | 24
  Occult Blood, BASELINE/DAY 1, 2+ | 1 | 1 | 0
  Occult Blood, BASELINE/DAY 1, 3+: number analyzed (Participants) | 54 | 37 | 24
  Occult Blood, BASELINE/DAY 1, 3+ | 4 | 0 | 1
  Occult Blood, ON IV TREATMENT/DAY 2, Trace: number analyzed (Participants) | 58 | 31 | 23
  Occult Blood, ON IV TREATMENT/DAY 2, Trace | 3 | 0 | 1
  Occult Blood, ON IV TREATMENT/DAY 2, 1+: number analyzed (Participants) | 58 | 31 | 23
  Occult Blood, ON IV TREATMENT/DAY 2, 1+ | 1 | 0 | 0
  Occult Blood, ON IV TREATMENT/DAY 2, 2+: number analyzed (Participants) | 58 | 31 | 23
  Occult Blood, ON IV TREATMENT/DAY 2, 2+ | 0 | 0 | 2
  Occult Blood, ON IV TREATMENT/DAY 2, 3+: number analyzed (Participants) | 58 | 31 | 23
  Occult Blood, ON IV TREATMENT/DAY 2, 3+ | 1 | 1 | 0
  Occult Blood, ON IV TREATMENT/DAY 3, Trace: number analyzed (Participants) | 32 | 20 | 9
  Occult Blood, ON IV TREATMENT/DAY 3, Trace | 0 | 1 | 0
  Occult Blood, ON IV TREATMENT/DAY 3, 3+: number analyzed (Participants) | 32 | 20 | 9
  Occult Blood, ON IV TREATMENT/DAY 3, 3+ | 0 | 0 | 1
  Occult Blood, ON IV TREATMENT/DAY 5, Trace: number analyzed (Participants) | 13 | 6 | 0
  Occult Blood, ON IV TREATMENT/DAY 5, Trace | 2 | 0 |
  Occult Blood, ON IV TREATMENT/DAY 7, Trace: number analyzed (Participants) | 4 | 1 | 0
  Occult Blood, ON IV TREATMENT/DAY 7, Trace | 1 | 0 |
  Occult Blood, ORAL - FIRST DAY, Trace: number analyzed (Participants) | 51 | 31 | 22
  Occult Blood, ORAL - FIRST DAY, Trace | 2 | 1 | 1
  Occult Blood, ORAL - FIRST DAY, 1+: number analyzed (Participants) | 51 | 31 | 22
  Occult Blood, ORAL - FIRST DAY, 1+ | 3 | 1 | 0
  Occult Blood, ORAL - FIRST DAY, 2+: number analyzed (Participants) | 51 | 31 | 22
  Occult Blood, ORAL - FIRST DAY, 2+ | 1 | 0 | 0
  Occult Blood, ORAL - FIRST DAY, 3+: number analyzed (Participants) | 51 | 31 | 22
  Occult Blood, ORAL - FIRST DAY, 3+ | 0 | 1 | 0
  Occult Blood, ORAL - DAY 7-10, Trace: number analyzed (Participants) | 45 | 30 | 22
  Occult Blood, ORAL - DAY 7-10, Trace | 1 | 0 | 1
  Occult Blood, ORAL - DAY 7-10, 2+: number analyzed (Participants) | 45 | 30 | 22
  Occult Blood, ORAL - DAY 7-10, 2+ | 1 | 0 | 1
  Occult Blood, ORAL - DAY 7-10, 3+: number analyzed (Participants) | 45 | 30 | 22
  Occult Blood, ORAL - DAY 7-10, 3+ | 0 | 0 | 1
  Occult Blood, POST THERAPY DAY 12-18, Trace: number analyzed (Participants) | 53 | 32 | 22
  Occult Blood, POST THERAPY DAY 12-18, Trace | 1 | 1 | 1
  Occult Blood, POST THERAPY DAY 12-18, 1+: number analyzed (Participants) | 53 | 32 | 22
  Occult Blood, POST THERAPY DAY 12-18, 1+ | 1 | 1 | 0
  Occult Blood, POST THERAPY DAY 12-18, 2+: number analyzed (Participants) | 53 | 32 | 22
  Occult Blood, POST THERAPY DAY 12-18, 2+ | 1 | 1 | 0
  Occult Blood, POST THERAPY DAY 12-18, 3+: number analyzed (Participants) | 53 | 32 | 22
  Occult Blood, POST THERAPY DAY 12-18, 3+ | 1 | 0 | 1
  Protein, BASELINE/DAY 1, Trace: number analyzed (Participants) | 54 | 37 | 24
  Protein, BASELINE/DAY 1, Trace | 7 | 5 | 5
  Protein, BASELINE/DAY 1, 1+: number analyzed (Participants) | 54 | 37 | 24
  Protein, BASELINE/DAY 1, 1+ | 6 | 4 | 5
  Protein, BASELINE/DAY 1, 2+: number analyzed (Participants) | 54 | 37 | 24
  Protein, BASELINE/DAY 1, 2+ | 1 | 0 | 1
  Protein, BASELINE/DAY 1, 3+: number analyzed (Participants) | 54 | 37 | 24
  Protein, BASELINE/DAY 1, 3+ | 1 | 0 | 0
  Protein, ON IV TREATMENT/DAY 2, Trace: number analyzed (Participants) | 58 | 31 | 23
  Protein, ON IV TREATMENT/DAY 2, Trace | 4 | 6 | 4
  Protein, ON IV TREATMENT/DAY 2, 1+: number analyzed (Participants) | 58 | 31 | 23
  Protein, ON IV TREATMENT/DAY 2, 1+ | 7 | 7 | 4
  Protein, ON IV TREATMENT/DAY 3, Trace: number analyzed (Participants) | 32 | 20 | 9
  Protein, ON IV TREATMENT/DAY 3, Trace | 4 | 3 | 0
  Protein, ON IV TREATMENT/DAY 3, 1+: number analyzed (Participants) | 32 | 20 | 9
  Protein, ON IV TREATMENT/DAY 3, 1+ | 3 | 2 | 3
  Protein, ON IV TREATMENT/DAY 3, 2+: number analyzed (Participants) | 32 | 20 | 9
  Protein, ON IV TREATMENT/DAY 3, 2+ | 1 | 0 | 0
  Protein, ON IV TREATMENT/DAY 5, Trace: number analyzed (Participants) | 13 | 6 | 0
  Protein, ON IV TREATMENT/DAY 5, Trace | 2 | 0 |
  Protein, ON IV TREATMENT/DAY 5, 1+: number analyzed (Participants) | 13 | 6 | 0
  Protein, ON IV TREATMENT/DAY 5, 1+ | 0 | 1 |
  Protein, ORAL - FIRST DAY, Trace: number analyzed (Participants) | 51 | 31 | 22
  Protein, ORAL - FIRST DAY, Trace | 2 | 3 | 1
  Protein, ORAL - FIRST DAY, 1+: number analyzed (Participants) | 51 | 31 | 22
  Protein, ORAL - FIRST DAY, 1+ | 0 | 4 | 2
  Protein, ORAL - FIRST DAY, 2+: number analyzed (Participants) | 51 | 31 | 22
  Protein, ORAL - FIRST DAY, 2+ | 1 | 0 | 0
  Protein, ORAL - DAY 7-10, Trace: number analyzed (Participants) | 45 | 30 | 22
  Protein, ORAL - DAY 7-10, Trace | 7 | 4 | 6
  Protein, ORAL - DAY 7-10, 1+: number analyzed (Participants) | 45 | 30 | 22
  Protein, ORAL - DAY 7-10, 1+ | 6 | 5 | 4
  Protein, ORAL - DAY 7-10, 2+: number analyzed (Participants) | 45 | 30 | 22
  Protein, ORAL - DAY 7-10, 2+ | 1 | 1 | 1
  Protein, POST THERAPY DAY 12-18, Trace: number analyzed (Participants) | 53 | 32 | 22
  Protein, POST THERAPY DAY 12-18, Trace | 8 | 6 | 2
  Protein, POST THERAPY DAY 12-18, 1+: number analyzed (Participants) | 53 | 32 | 22
  Protein, POST THERAPY DAY 12-18, 1+ | 3 | 4 | 3
  Protein, POST THERAPY DAY 12-18, 2+: number analyzed (Participants) | 53 | 32 | 22
  Protein, POST THERAPY DAY 12-18, 2+ | 0 | 1 | 0
  pH, Post-Baseline Maximum, 8.5: number analyzed (Participants) | 57 | 35 | 25
  pH, Post-Baseline Maximum, 8.5 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected up to follow-up (Day 28).
Description: Safety population was used.
Arm/Group | Gepotidacin 750 mg q12h | Gepotidacin 1000 mg q12h | Gepotidacin 1000 mg q8h
All-Cause Mortality (participants affected / at risk) | 0/58 | 1/39 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/39 | 0/25
Other Adverse Events (participants affected / at risk) | 30/58 | 20/39 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gepotidacin 750 mg q12h (N=58) | Gepotidacin 1000 mg q12h (N=39) | Gepotidacin 1000 mg q8h (N=25)
Cellulitis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gepotidacin 750 mg q12h (N=58) | Gepotidacin 1000 mg q12h (N=39) | Gepotidacin 1000 mg q8h (N=25)
Nausea (Gastrointestinal disorders) | 12 | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 5
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3
Flatulence (Gastrointestinal disorders) | 3 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 3 | 0
Headache (Nervous system disorders) | 6 | 1 | 0
Infusion site extravasation (General disorders) | 3 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.